

# STATISTICAL ANALYSIS PLAN

### STUDY TITLE:

An Open-label, Single-center, Three-part Study in Healthy Subjects to Investigate the Effect of Givinostat on the Pharmacokinetics of Midazolam and Dabigatran, the Effect of Clarithromycin on the Pharmacokinetics of Givinostat and the Pharmacokinetics of Single and Multiple Doses of Givinostat.

Protocol Code: ITF/2357/55

Type: Interventional, Pharmacokinetic and Drug-Drug Interaction

Trial

EudraCT No.: 2021-005756-11

Version: 1.0

Date of SAP: 24MAR2022

Supersedes Version: None

Date of Superseded Version: Not applicable

Sponsor: ITALFARMACO S.p.A

Via dei Lavoratori, 54

20092 Cinisello Balsamo (MI), Italy

with its registered office at Viale Fulvio Testi, 330,

Milan (MI), Italy www.italfarmaco.com Phone: + 39 02 64431 Fax: + 39 02 644346

Clinical Pharmacology Unit: PPD

### CONFIDENTIALITY DISCLAIMER

This document is confidential and is available for review to investigators, regulatory bodies and study audit personnel. No part of this document may be used, published, copied or otherwise disclosed without prior written authorization from PPD

or the Sponsor of this study.



Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 1. SIGNATURE PAGE

# 1.1. Clinical Research Unit





# 2. CONTENTS AND ABBREVIATIONS

# 2.1. Table of Contents

| 1. | SIGNATURE PAGE | 2 |
|---|---|---|
| | 1.1. CLINICAL RESEARCH UNIT | 2 |
| | 1.2. SPONSOR'S REPRESENTATIVE | 2 |
| 2. | CONTENTS AND ABBREVIATIONS | 3 |
| | 2.1. TABLE OF CONTENTS | 3 |
| | 2.2. LIST OF ABBREVIATIONS | |
| 3. | INTRODUCTION | 8 |
| 4. | STUDY OBJECTIVES | 8 |
| | 4.1. PRIMARY | 8 |
| | 4.2. SECONDARY | |
| 5. | INVESTIGATIONAL PLAN | 8 |
| | 5.1. STUDY DESIGN | 8 |
| | 5.1.1. Rational for Study Design. | |
| | 5.2. STUDY PLAN | |
| | 5.2.1. Part 3 - Pharmacokinetics of Givinostat and its Metabolites Fo | |
| | and Multiple Oral Doses of Givinostat | |
| | 5.3. NUMBER OF PARTICIPANTS AND SAMPLE SIZE ESTIMATION | 9 |
| | 5.3.1. Part 3 | 10 |
| | 5.4. RANDOMIZATION | 10 |
| | 5.5. BLINDING | 10 |
| 5. | STUDY ASSESSMENTS | 10 |
| | 6.1. SAFETY ASSESSMENTS | 10 |
| | 6.1.1. Medical History | 10 |
| | 6.1.2. Physical Examination | 11 |
| | 6.1.3. Weight, Height and Body Mass Index | <i>11</i> |
| | 6.1.4. Vital Signs | 11 |
| | 6.1.5. 12 Lead Electrocardiogram | 11 |
| | 6.1.6. Laboratory Safety Tests | 11 |
| | 6.1.7. Adverse Events | |
| | 6.1.8. Previous and Concomitant Medications | 14 |
| | 6.2. PHARMACOKINETIC ASSESSMENTS | 14 |
| | 6.2.1. Blood Sampling for Pharmacokinetic Assessments | |
| | 6.2.2. Urine Sampling for Pharmacokinetic Assessments | |
| | 6.2.3. Plasma Pharmacokinetic Parameters | |
| | 6.2.4. Urinary Pharmacokinetic Parameters | 18 |
| 7. | STUDY ENDPOINTS | 18 |
| | 7.1. PRIMARY | 18 |
| | 7.2. SECONDARY | 18 |
| 2 | ANALYSIS POPULATIONS | 10 |

| | 8.1. PART 3 | 19 |
|---|---|---|
| | 8.1.1. Part 3 Safety Analysis Population | 19 |
| | 8.1.2. Part 3 Pharmacokinetic Analysis Population | 19 |
| 9. | DATA REVIEW / TRANSFORMATION | 20 |
| | 9.1. DATA MANAGEMENT | 20 |
| | 9.2. ACCEPTANCE OF DATA | 20 |
| | 9.3. DATA TRANSFORMATION (CDISC) | 20 |
| 10. | STATISTICAL METHODS | 22 |
| | 10.1. GENERAL CONSIDERATIONS | 23 |
| | 10.2. SUBJECTS' DISPOSITION | 23 |
| | 10.3. PROTOCOL DEVIATIONS | |
| | 10.4. PLASMA PHARMACOKINETIC CONCENTRATIONS | 23 |
| | 10.5. PLASMA PHARMACOKINETIC PARAMETERS | 24 |
| | 10.6. URINARY DATA | |
| | 10.7. URINARY PHARMACOKINETIC PARAMETERS | 25 |
| 11. | PRESENTATION OF RESULTS | 25 |
| | 11.1. STATISTICAL OUTPUT SPECIFICATION | 25 |
| | 11.2. PLANNED TABLES, FIGURES, AND SUBJECT DATA LISTINGS | 26 |
| | 11.2.1. In-text Tables and Figures | |
| | 11.2.2. Tables, Figures and Graphs Referred to But Not Included in the | |
| | 14 of CSR) | |
| | 11.2.3. List of Subject Data Listings (Section 16.2 of CSR) | 40 |
| 12. | REFERENCES | 49 |
| 13. | APPENDICES | 50 |
| | APPENDIX A. PLANNED TABLES, FIGURES, AND SUBJECT DATA LISTINGS | 50 |
| | A.1. In-text Tables and Figures – For CSR Synopsis | 50 |
| | A.2. In-text Tables and Figures – For CSR Body Text | 58 |
| | A.3. Tables, Figures and Graphs Referred to But Not Included in the Text of CSR) | |
| | A.4. List of Subject Data Listings (Section 16.2 of CSR) | |
| 14 | ANNEYES | |
| - | | 4 |

### 2.2. List of Abbreviations

α Type I Error (Significance Level)

Ab Antibody

ADaM Analysis Data Model

ADAMIG Analysis Data Model Implementation Guide
ADPC Analysis Data Pharmacokinetic Concentrations
ADPP Analysis Data Pharmacokinetic Parameters

ADSL Subject-Level Analysis

AE Adverse Event
ALP Alkaline Phosphatase
ALT Alanine Aminotransferase

Amean Arithmetic Mean ANOVA Analysis of Variance

aPTT Activated Partial Thromboplastin Time

AST Aspartate Aminotransferase ATC Anatomic Therapeutic Chemical

AUC Area Under the Concentration Versus Time Curve

AUC from Time Zero to Last Sampling Time with Quantifiable Concentrations

AUC<sub>0-∞</sub> AUC from Time Zero to Infinity

AUC 0-1,55 AUC Corresponding to the Dosing Interval, at Steady State

AURCo.t Area Under the Urinary Excretion Rate Curve from Time 0 to the Last Rate

%AUCextrap Residual Area or Percentage of Extrapolated Part of AUC₀∞

BDS Basic Data Structure

BLQ Below the Limit of Quantification

BMI Body Mass Index
bpm Beats Per Minute
Co Pre-dose Concentration
CI Confidence Interval
Cl Total Body Clearance
CK Creatine Kinase

Cl/F Total Body Clearance Affected by the Bioavailability Factor

Cl<sub>R</sub> Renal Clearance

Cl<sub>R</sub>/F Renal Clearance Affected by the Bioavailability Factor

C<sub>last</sub> Last Quantifiable Concentration
C<sub>max</sub> Maximum Observed Concentration

Cmax.55 Maximum Observed Plasma Concentration at Steady State

Crca Creatinine Clearance
CSP Clinical Study Protocol
CSR Clinical Study Report
CV% Coefficient of Variation
CYP Cytochrome P450
DBP Diastolic Blood Pressure
DDI Drug-Drug Interaction

DM Demographics
ECG Electrocardiogram
F Bioavailability Factor

FDA Food and Drug Administration GGT Gamma-Glutamyltransferase GLP Good Laboratory Practices ITF/2357/55 Version: 1.0 Date: 24MAR2022



Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

Gmesn Geometric Mean

GMR Geometric Least Square Means Ratio
GCV% Geometric Coefficient of Variation
GSD Geometric Standard Deviation

H<sub>0</sub> Null Hypothesis
H<sub>1</sub> Alternative Hypothesis
HBsAg Hepatitis B Surface Antigen
hCG Human Chorionic Gonadotropin
HCVAb Hepatitis C Virus Antibodies
HIV Human Immunodeficiency Virus

ICH International Conference on Harmonization

INR International Normalized Ratio
ISCV% Intra-Subject Coefficient of Variation

IV Intravenous

LC-MS/MS Liquid Chromatography with Tandem Mass Spectrometry

LDH Lactate Dehydrogenase

LLOQ Lower Limit of Quantification

LSmeans Least Square Means

MCH Mean Corpuscular Hemoglobin

MCHC Mean Corpuscular Hemoglobin Concentration

MCV Mean Corpuscular Volume

MedDRA Medical Dictionary for Regulatory Activities

MSE Mean Square Error MW Molecular Weight

NCA Non-Compartmental Analysis
PC Pharmacokinetic Concentrations
PCL Protocol Clarification Letter

P-gp P-Glycoprotein

PP Pharmacokinetic Parameters PT MedDRA Preferred Term

QTcF Corrected QT Interval by Fridericia

RBC Red Blood Cell

RDW-CV Coefficient Variation of the Red Cell Distribution Width
RSQ Goodness of Fit for the Terminal Elimination Phase

rtf Rich Text File

SAE Serious Adverse Event SAP Statistical Analysis Plan SAR Serious Adverse Reaction

SARS-CoV-2 Severe Acute Respiratory Syndrome Coronavirus 2

SAS Statistical Analysis Software SBP Systolic Blood Pressure SD Standard Deviation

SDTM Study Data Tabulation Model

SDTMIG Study Data Tabulation Model Implementation Guide

SOC MedDRA System Organ Class SOP Standard Operating Procedure TEAE Treatment-Emergent Adverse Events

TFLs Tables, Figures and Listings

T<sub>max</sub> Time to Maximum Observed Concentration

T<sub>max,ss</sub> Time to Maximum Observed Concentration at Steady State

ITF/2357/55 Version: 1.0 Date: 24MAR2022



Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

| TOST | Two One-Sided T-Tests |
|------|-----------------------------|
| TSH | Thyroid-Stimulating Hormone |
| to | Time of Dosing (t=0h) |

t<sub>½</sub> Apparent Terminal Elimination Half-Life

ULOQ Upper Limit of Quantification V<sub>D</sub> Apparent Volume of Distribution

V<sub>D</sub>/F Apparent Volume of Distribution Affected by the Bioavailability Factor (F)

WBC White Blood Cell

WHO World Health Organization

λ<sub>z</sub> Apparent Terminal Elimination Rate Constant

τ Dosing Interval

Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 3. INTRODUCTION

This Statistical Analysis Plan (SAP) details the statistical methodology to be used in analysing study data and outlines the statistical programming specifications for the Tables, Figures and Listings (TFLs). This document describes the variables and populations, anticipated data transformation and manipulations and other details of the analysis not provided in the Clinical Study Protocol (CSP).

The described analyses are based on the final CSP version 1.0, dated 29NOV2021 [1] and a Protocol Clarification Letter (PCL) dated 25FEB2022. This SAP was finalized prior to data base lock and conduct of the statistical analyses. For each part of the study at the time of the Blind Review Process, a Data Blind Review Process Minute will be prepared and attached to this document (Annex 5).

Additional pharmacokinetic and statistical analysis may be performed to supplement the planned analyses described in this SAP. These supplemental analyses will be identified and presented in the Clinical Study Report (CSR).

### 4. STUDY OBJECTIVES

### 4.1. Primary

 To evaluate the plasma and urine pharmacokinetics of givinostat and its metabolites following single and multiple oral doses of givinostat (Part 3).

# 4.2. Secondary

To assess the safety and tolerability of single and multiple doses of givinostat (Part 3).

# 5. INVESTIGATIONAL PLAN

### 5.1. Study Design

This is a phase I, open-label, 3-part, fixed-sequence, non-randomized study in healthy male and female subjects.

Study parts may be conducted concomitantly.

# 5.1.1. Rational for Study Design

The rational for study design detailed in the CSP [1].

In Part 3, the pharmacokinetics of givinostat and its metabolites in plasma and urine following single- and multiple-doses of givinostat will be investigated.

# 5.2. Study Plan

# 5.2.1. Part 3 – Pharmacokinetics of Givinostat and its Metabolites Following Single and Multiple Oral Doses of Givinostat

Subjects will be confined in PPD from Day -1 to Day 17.

On Day 1 and Day 13, givinostat 50 mg as oral suspension will be administered as a single dose, in the morning, following an overnight fasting of at least 8 hours and subjects will remain fasted until at least 4 hours post dose. No fluids will be allowed from 1 hour before dosing until 2 hours post dose. Water will be provided ad libitum at all other times.

From Day 5 to Day 12, subjects will receive givinostat 50 mg as oral suspension, twice a day, in the morning and in the evening. On Days 1 and 13, givinostat will be administered with the subjects in a semi-recumbent position and will remain semi-recumbent until at least 4 hours post-dose.

The following assessments will be performed:

- Blood collection for pharmacokinetic analysis on Days 1 to 5 and 9 to 17.
- Urine collection for pharmacokinetic analysis on Days 1 to 5 and 13 to 17 (Baseline urine collection is on day -1).
- Vital signs measurements (BP, PR and RR) on Days 1 and 5 to 13.
- 12-lead ECG on Days 1 and 4 to 13.
- Blood collection for laboratory tests (hematology and biochemistry on Day 9 and hematology on Days 6 and 13).

Subjects will be discharged from PPD on the morning of Day 17 if allowed by the investigator based on their medical condition. The following procedures will be performed:

- Physical examination.
- Collection of body weight.
- Vital signs measurements (BP, PR, RR and body temperature).
- 12-lead ECG.
- Safety laboratory assessments (hematology, biochemistry, coagulation and urinalysis).
- Serum pregnancy test for all female subjects.

Subjects will return to PPD 10 to 14 days after the end of study to undergo additional assessments as required as per protocol.

The total duration of Part 3 for each subject will be up to approximately 8 weeks from Screening to Follow-up visit, divided as follows:

- Screening: up to 21 days
- Treatment Period: Days 1 to 17
- Safety follow-up visit: 12±2 days

### 5.3. Number of Participants and Sample Size Estimation

To ensure enough subjects with evaluable data complete each study part, a total of fifty-four (54) healthy male and female subjects are planned to be enrolled as follows:

- Part 1: twenty-six (26) subjects
- Part 2: twenty (20) subjects

# 5.2. Study Plan

# 5.2.1. Part 3 – Pharmacokinetics of Givinostat and its Metabolites Following Single and Multiple Oral Doses of Givinostat

Subjects will be confined in PPD from Day -1 to Day 17.

On Day 1 and Day 13, givinostat 50 mg as oral suspension will be administered as a single dose, in the morning, following an overnight fasting of at least 8 hours and subjects will remain fasted until at least 4 hours post dose. No fluids will be allowed from 1 hour before dosing until 2 hours post dose. Water will be provided ad libitum at all other times.

From Day 5 to Day 12, subjects will receive givinostat 50 mg as oral suspension, twice a day, in the morning and in the evening. On Days 1 and 13, givinostat will be administered with the subjects in a semi-recumbent position and will remain semi-recumbent until at least 4 hours post-dose.

The following assessments will be performed:

- Blood collection for pharmacokinetic analysis on Days 1 to 5 and 9 to 17.
- Urine collection for pharmacokinetic analysis on Days 1 to 5 and 13 to 17 (Baseline urine collection is on day -1).
- Vital signs measurements (BP, PR and RR) on Days 1 and 5 to 13.
- 12-lead ECG on Days 1 and 4 to 13.
- Blood collection for laboratory tests (hematology and biochemistry on Day 9 and hematology on Days 6 and 13).

Subjects will be discharged from PPD on the morning of Day 17 if allowed by the investigator based on their medical condition. The following procedures will be performed:

- Physical examination.
- Collection of body weight.
- Vital signs measurements (BP, PR, RR and body temperature).
- 12-lead ECG.
- Safety laboratory assessments (hematology, biochemistry, coagulation and urinalysis).
- Serum pregnancy test for all female subjects.

Subjects will return to PPD 10 to 14 days after the end of study to undergo additional assessments as required as per protocol.

The total duration of Part 3 for each subject will be up to approximately 8 weeks from Screening to Follow-up visit, divided as follows:

- Screening: up to 21 days
- Treatment Period: Days 1 to 17
- Safety follow-up visit: 12±2 days

### 5.3. Number of Participants and Sample Size Estimation

To ensure enough subjects with evaluable data complete each study part, a total of fifty-four (54) healthy male and female subjects are planned to be enrolled as follows:

- Part 1: twenty-six (26) subjects
- Part 2: twenty (20) subjects

Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- Part 3: eight (8) subjects

Each subject will participate in one study part only.

### 5.3.1. Part 3

A sample size of 8 subjects will be enrolled. The sample size was determined by practical considerations and not based on statistical power calculations.

### 5.4. Randomization

This is a fixed sequence study. Randomization is not applicable.

# 5.5. Blinding

The study will be conducted as open label. Blinding procedures are not applicable.

### 6. STUDY ASSESSMENTS

For each study part, a summary of procedures for study assessments are presented in Section 2 of the CSP (Study Flow-Chart and Study Design Diagram) [1].

# 6.1. Safety Assessments

Subjects' safety will be monitored during the study.

Safety assessments will include pre-study medical history, physical examination, vital signs, 12-lead ECG, clinical laboratory tests and adverse event (AE) monitoring. Additional safety measurements may be performed at the discretion of the investigator for reasons related to subject safety.

Medications will be mentioned according to the World Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) classification system.

# 6.1.1. Medical History

Medical history will cover all relevant past or present information related to subject's health at the time of informed consent signature.

Medical history at screening will include past or present relevant cardiovascular, respiratory, renal, genitourinary, gastrointestinal, hepatic, hematological, immunological, endocrine, dermatological, musculoskeletal, neurological, psychiatric, drug and surgical history, or any other diseases or disorders.

Medical history will be referred in accordance with the Medical Dictionary for Regulatory Activities (MedDRA), version 24.1 or higher.

Adverse events related to medical history will be identified.

# 6.1.2. Physical Examination

Physical examination at screening and end-of-study will include: general appearance; skin; head and neck; thorax and abdomen; pulmonary auscultation; cardiac auscultation; abdomen palpation; limbs; brief neurological examination.

# 6.1.3. Weight, Height and Body Mass Index

The body height and weight values as well as the body mass index (BMI) will be recorded in the electronic case report form (eCRF) and will be determined at Screening. Only body weight will be determined also at admission and end-of-study.

The subjects' body weight will preferably be measured using the same weighing scale for all subjects and throughout the study. The weighing scale should have a precision of at least 0.5 kg.

### 6.1.4. Vital Signs

Vital signs will include:

- Systolic blood pressure (SBP).
- Diastolic blood pressure (DBP).
- Pulse rate (PR).
- Respiratory rate (RR).
- Body temperature.

# 6.1.5. 12 Lead Electrocardiogram

A 12-lead ECG will be performed preferably before the blood collection. The corrected QT interval by Fridericia (QTcF) will be analyzed.

# 6.1.6. Laboratory Safety Tests

The following laboratory parameters will be tested:

- Hematology:
  - Red blood cell (RBC) count.
  - White blood cell (WBC) count.
  - WBC differential count:
    - Neutrophils.
    - Eosinophils.
    - Basophils.
    - Lymphocytes.
    - Monocytes.
  - Hemoglobin.
  - Mean corpuscular volume (MCV).
  - Mean corpuscular hemoglobin (MCH).
  - Mean corpuscular hemoglobin concentration (MCHC).
  - Coefficient variation of the red cell distribution width (RDW-CV).
  - Hematocrit.
  - Platelet count.
  - Mean platelet volume.

- Coagulation:
  - Prothrombin rate.
  - Prothrombin time.
  - Prothrombin time international normalized ratio (INR).
  - Activated partial thromboplastin time (aPTT).
- General biochemistry:
  - Total bilirubin.
  - Direct bilirubin.
  - Indirect bilirubin.
  - Alkaline phosphatase (ALP).
  - Amylase.
  - Aspartate aminotransferase (AST).
  - Alanine aminotransferase (ALT).
  - Lactate dehydrogenase (LDH).
  - Cystatin C.
  - C-reactive protein.
  - Gamma-glutamyltransferase (GGT).
  - Creatinine kinase (CK).
  - Total protein.
  - Albumin.
  - Uric acid.
  - Triglycerides.
  - Total cholesterol.
  - Low-density lipoprotein-cholesterol (LDL-C).
  - High-density lipoprotein-cholesterol (HDL-C).
  - Sodium.
  - Potassium
  - Chloride.
  - Calcium.
  - Magnesium.
  - Glucose.
  - Creatinine.
  - Urea.
  - Thyroid-stimulating hormone (TSH).
  - Estimated creatinine clearance (CrcL).
- Viral Serology:
  - Human Immunodeficiency Virus (HIV):
    - HIV-1 (anti-HIV-1Ab).
    - HIV-2 (anti-HIV-2Ab).
  - Hepatitis B (HBsAg)
  - Hepatitis C (anti-HCVAb).
- Beta-human chorionic gonadotropin (beta-hCG) pregnancy tests:
  - Serum.
  - Urine.
- Urinalysis:
  - pH.

- Specific gravity.
- Protein.
- Hemoglobin.
- Glucose.
- Ketones.
- Bilimbin
- Nitrites.
- Urobilinogen.
- Microscopy.
- Drugs-of-abuse urine test:
  - Cannabinoids.
  - Opiates.
  - Cocaine.
  - Amphetamines.
  - Benzodiazepines.
- Ethanol urine test.
- Cotinine urine test.
- Follicle-stimulating hormone (FSH) test.
- Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) diagnostic tests.

# 6.1.7. Adverse Events

The occurrence of clinical AEs will be monitored throughout the study.

Clinically significant abnormalities in laboratory safety tests, vital signs and physical examination will be reported as AEs.

Treatment-emergent AEs (TEAEs) are defined as AEs not present prior to first administration of investigational product, or AEs present before first administration of investigational product that worsen after the subject receives the first dose of investigational product. TEAEs that occur after administration of investigational product during the washout of a given period will be assigned to the treatment administered in that period.

The following information will be used for the description of the AEs:

- Reported Term.
- Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) coding.
- MedDRA Preferred Term (PT) coding.
- Start date and time.
- End date and time.
- Seriousness.
- Severity:
  - Mild
  - Moderate.
  - Severe.
- Relationship (causality) for each treatment administrated, per part.
  - Reasonably Possible.
  - Not Reasonably Possible.
  - Unknown.

- Action taken:
  - Dose Increased
  - Dose Not Changed.
  - Dose Rate Reduced.
  - Dose Reduced.
  - Drug Interrupted.
  - Drug Withdrawn.
  - Not Applicable.
  - Unknown.
- Concomitant medication.
- Outcome:
  - Fatal.
  - Not Recovered / Not Resolved.
  - Recovered / Resolved.
  - Recovered / Resolved with Sequelae.
  - Recovering / Resolving.
  - Unknown.
- Most recent study treatment taken.
- Last dosing date.

### 6.1.8. Previous and Concomitant Medications

A previous medication is any medication for which the end date is prior to first dosing. A concomitant medication is any medication ongoing or initiated after first dosing.

For all study parts, the use of any medications including Over-the-Counter (OTC) products (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) is forbidden from 28 days or within 5 half-lives of the medicinal product, whichever is longer, prior to admission up to last sample for pharmacokinetics assessment, except for medications for the treatment of AEs.

Any medication (previous or concomitant) taken within the period of medication restriction must be recorded in the eCRF. If concomitant medication is ongoing at the follow-up visit, no end date will be provided in the eCRF.

For each study part, previous and concomitant medications used by study participants during the study and their judged impact on the pharmacokinetic assessment will be listed in the respective Data Blind Review Meeting/ Process Minute (Annex 5).

Concomitant medications will be coded according to the WHO ATC classification system.

### 6.2. Pharmacokinetic Assessments

# 6.2.1. Blood Sampling for Pharmacokinetic Assessments

In each study part, while subject is confined at the clinical research unit, blood samples will be taken preferably via an indwelling cannula placed in a vein of an upper limb of the subject. During ambulatory visits, blood samples will be taken by direct venipuncture.

The actual time of all pharmacokinetic blood draws will be recorded and reported for all subjects. The pre-dose blood sample will be collected within 30 minutes before dosing. The post-dose blood samples will be collected within ±3 minutes from the scheduled sampling time. Greater deviations will be reported as a protocol deviation and its cause will be recorded.

In case blood sampling for pharmacokinetics and other procedures coincide in time, blood draws will have priority unless other procedures are necessary for assuring subject's safety.

will carry out the determination of plasma levels of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563), midazolam, 1-hydroxymidazolam and total and free dabigatran in accordance with the applicable principles of Good Laboratory Practices (GLP), using a previously validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) analytical method.

The planned lower limit of quantification (LLOQ) and upper limit of quantification (ULOQ) for:

- givinostat are 1 and 100 ng/mL.
- givinostat metabolite ITF2374 are 1 and 100 ng/mL.
- givinostat metabolite ITF2375 are 1 and 100 ng/mL.
- givinostat metabolite ITF2440 are 10 and 500 ng/mL.
- givinostat metabolite ITF2563 are 2 and 125 ng/mL.
- midazolam are 100 and 100000 pg/mL.
- 1-hydroxymidazolam are 100 and 50000 pg/mL.
- total dabigatran are 1 and 400 ng/mL.
- free dabigatran are 1 and 400 ng/mL.

LLOQ represents a value lower than or equal to 1/20 of estimated C<sub>max</sub> value. Any adjustment to this range will be documented in the study specific Bioanalytical Report, which will supersede the indicated range.

### 6.2.1.1. Part 3

A total of forty-eight (48) blood samples will be collected as follows:

- Twenty-two (22) blood samples of 6 mL each will be collected in sodium heparin tubes at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours after the administration of givinostat, on Days 1 and 13, for the determination of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) plasma concentrations.
- Four (4) blood samples of 6 mL each will be collected in sodium heparin tubes before the morning dose of givinostat on Days 9, 10, 11 and 12, for the determination of pre-dose (Ctrough) plasma concentration of givinostat and metabolites.

### 6.2.2. Urine Sampling for Pharmacokinetic Assessments

### 6.2.2.1. Part 3

Urine will be collected on Day -1 (baseline) and in the following intervals, on Days 1 and 13, for the determination of the amounts of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) excreted in urine: 0-12, 12-24, 24-36, 36-48, 48-72 and 72-96 post-dose.

The date and actual time of urine collection start and completion will be recorded and reported for all subjects.

will carry out the determination of urine levels of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) in accordance with the applicable principles of GLP using a previously validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) analytical method.

The planned lower limit of quantification (LLOQ) and upper limit of quantification (ULOQ) for:

- givinostat are 10 and 2500 ng/mL.
- givinostat metabolite ITF2374 are 5 and 2500 ng/mL.
- givinostat metabolite ITF2375 are 4 and 800 ng/mL.
- givinostat metabolite ITF2440 are 150 and 25000 ng/mL.
- givinostat metabolite ITF2563 are 10 and 5000 ng/mL.

### 6.2.3. Plasma Pharmacokinetic Parameters

The following pharmacokinetic parameters will be derived by standard non-compartmental analysis (NCA) methods from the single-dose plasma concentration versus time profiles, for:

- Part 3 (Day 1):
  - givinostat.
  - givinostat metabolites (ITF2374, ITF2375, ITF2440 and ITF2563).

| Parameter | Description |
|---|---|
| Cmax | Maximum observed concentration, directly obtained from the observed concentration versus time profile. |
| $T_{max}$ | Time of occurrence of maximum observed concentration. |
| AUC <sub>0-t</sub> <sup>1</sup> | Area under the concentration <i>versus</i> time curve (AUC) from time of dosing (t=0h) to the time of the last measurable concentration (t <sub>last</sub> ), calculated by the linear-up/log-down trapezoidal method. |
| AUC <sub>0-∞</sub> | Total AUC extrapolated to infinity, calculated as $AUC_{0-t} + \frac{c_{last}}{\lambda_z}$ , where $C_{last}$ |
| | is the last measurable concentration and $\lambda_z$ is the apparent terminal elimination rate constant. |
| %AUC <sub>extrap</sub> | Percentage of AUC <sub>0-∞</sub> due to extrapolation from the time of the last measurable concentration ( $t_{last}$ ) to infinity, i.e., residual area, calculated as $100 \cdot \frac{AUC_{0-\infty} - AUC_{0-t}}{AUC_{0-\infty}}$ . |
| $\lambda_z$ | Apparent first order elimination rate constant associated with the terminal (log-linear) portion of the concentration <i>versus</i> time curve. The parameter is estimated by linear least square regression analysis using the last three (or more) non-zero concentrations. |
| t <sub>1/2</sub> | Apparent terminal elimination half-life, calculated as $\frac{ln(2)}{\lambda_2}$ . |

In Part 3, for givinostat and its metabolites the last sampling time corresponds to 96 hours.

The upper and the lower timepoints and the number of timepoints used for  $\lambda_z$  estimation, as well as the goodness of fit for the terminal elimination phase (RSQ), will be reported. No values of  $\lambda_z$ , AUC<sub>0-∞</sub>, %AUC<sub>extrap</sub> and  $t_{4z}$  will be reported for cases where  $\lambda_z$  cannot be reliably determined.

The following pharmacokinetic parameters will be derived by standard NCA methods from the multiple-dose plasma concentration *varsus* time profiles, for:

# Part 3 (Day 13):

- givinostat.
- givinostat metabolites (ITF2374, ITF2375, ITF2440 and ITF2563).

| Parameter | Description |
|---|---|
| $C_{max,ss}$ | Maximum observed plasma concentration at steady state, directly obtained from the observed concentration versus time profile. |
| T <sub>max,55</sub> | Time of occurrence of maximum observed plasma concentration at steady state. |
| AUC <sub>0-T,SS</sub> | Area under the plasma concentration versus time curve corresponding to dosing interval, i.e., 12 hours, after steady state has been reached. This parameter is calculated by the linear-up/log-down trapezoidal method. |
| AUC <sub>0-t</sub> | AUC from time of dosing (t=0h) to the time of the last measurable concentration (t <sub>last</sub> ), calculated by the linear-up/log-down trapezoidal method. |
| $AUC_{0-\infty}$ | Total AUC extrapolated to infinity, calculated as $AUC_{0-t} + \frac{c_{last}}{\lambda_{-}}$ , where $C_{last}$ |
| | is the last measurable concentration and $\lambda_z$ is the apparent terminal elimination rate constant. |
| $\lambda_z$ | Apparent first order elimination rate constant associated with the terminal (log-linear) portion of the concentration <i>versus</i> time curve. The parameter is estimated by linear least square regression analysis using the last three (or more) non-zero concentrations. |
| t <sub>1/2</sub> | Apparent terminal elimination half-life, calculated as $\frac{ln(2)}{\lambda_z}$ . |
| CL <sub>ss</sub> /F | Apparent total body clearance affected by the bioavailability factor (F), calculated as $\frac{Dose}{AUC_{0-T,SS}}$ . |
| V <sub>D</sub> /F | Apparent volume of distribution affected by F, calculated as $\frac{Dose}{\lambda_z \cdot AUC_{0-T,88}}$ . |

The upper and the lower timepoints and the number of timepoints used for  $\lambda_z$  estimation, as well as the RSQ, will be reported.

No values of  $\lambda_z$ , AUC<sub>0-∞</sub>, %AUC<sub>extrap</sub> and  $t_{1/2}$  will be reported for cases where  $\lambda_z$  cannot be reliably determined.

For each study part, pharmacokinetic parameters will be estimated from the plasma concentration versus time profiles for all subjects in each pharmacokinetic analysis population.

Actual sampling times will be used for the pharmacokinetic analysis. All calculations will be performed using raw data.

In estimating the pharmacokinetic parameters, concentrations below the LLOQ before  $T_{max}$  will be set to zero. After Tmax, concentrations below the LLOQ will be considered as missing. However, in case of two or more consecutive concentrations below the LLOQ, the first value will be replaced by 1/2 of the LLOQ value and the next values will be considered as missing.

Additional pharmacokinetic parameters may be calculated for the plasma concentration versus time profiles, if considered appropriate and justified at the time of the pharmacokinetic analysis.

#### 6.2.4. Urinary Pharmacokinetic Parameters

The following pharmacokinetic parameters will be derived by standard NCA methods from the urine excretion profiles, for the first dose (Day 1, single-dose) and the last dose (Day 13, multiple-dose):

- Part 3:
  - givinostat.
  - givinostat metabolites (ITF2374, ITF2375, ITF2440 and ITF2563).

| Parameter | Description |
|-----------|-------------|

Maximum observed urinary excretion rate. Rmax

Time of occurrence of maximum urinary excretion rate. tumax Cumulative amount of drug excreted in urine, calculated as Amtcum

 $\sum$ (Concentration · Volume)

AURC0-t Area under the urine excretion rate curve from time zero to last measurable

observed excretion rate.

REC% Percentage of drug recovered in urine, calculated for givinostat as 100 ·

Amt<sub>CUM</sub>, and for givinostat metabolites as 100 ·

AMT CUM, Metabolie / MW Metabolite, where MW represents the molecular weight

DoseGivinostat/MWGivinostat

of the analyte.

Note: For givinostat, MW is 421.49 g/mol; for ITF2374, MW is 405.49 g/mol; for ITF2375, MW is 406.47 g/mol; for ITF2440, MW is 257.33

g/mol; and for ITF2563, MW is 178.19 g/mol.

Apparent renal clearance affected by F, calculated as Dose CLR/F

#### 7. STUDY ENDPOINTS

#### 7.1. Primary

 Givinostat and its metabolites plasma and urine concentrations and thereof derived pharmacokinetic parameters following single and multiple oral doses of givinostat (Part 3).

#### 7.2. Secondary

 Incidence and severity of AEs; changes in vital signs, physical examination, ECG and clinical laboratory tests following administration of single- and multiple-doses of givinostat (Part 3).

### 8. ANALYSIS POPULATIONS

The analysis populations are defined in accordance with the CSP [1].

For each study part, the subjects to be included in each analysis population will be reported in the respective Data Blind Review Process Minute (Annex 5).

For each study part, explanation of the reasons for exclusion of subjects from any analysis population will be provided in the respective Data Blind Review Process Minute (Annex 5) and in the CSR.

The list of subjects who complete each study part will be presented in Annex 6.

### 8.1. Part 3

# 8.1.1. Part 3 Safety Analysis Population

All subjects who receive at least one dose of the IMP in Part 3 of the study will constitute the Part 3 Safety Analysis Population.

Part 3 safety data analysis will be performed for all subjects in the Part 3 Safety Analysis Population.

### 8.1.2. Part 3 Pharmacokinetic Analysis Population

### 8.1.2.1. Part 3 Single-Dose Pharmacokinetic Analysis Population

Part 3 Single-Dose Pharmacokinetic Analysis Population will include all subjects enrolled in Part 3 of the study, who are expected to provide evaluable pharmacokinetic data for the givinostat single-dose administration (Day 1), without deviations affecting pharmacokinetic interpretation.

The following reasons justify the exclusion of the pharmacokinetic data of a subject from the Part 3 single-dose pharmacokinetic analysis population:

 Protocol violation considered to have a potentially relevant effect on the pharmacokinetic results of the study.

NOTE: These protocol violations will be reported in the Data Blind Review Process Minute (Annex 5), and their impact will be assessed at the time of pharmacokinetic analysis.

Subject experienced vomiting or diarrhea.

NOTE: Subjects that experienced vomiting or diarrhoea during this study part will be reported in the Data Blind Review Process Minute (Annex 5), and their exclusion will be assessed at the time of pharmacokinetic analysis.

- Subject with pre-dose concentration > 5% of the C<sub>max</sub> value of the corresponding pharmacokinetic profile.
  - NOTE: This exclusion will be assessed at the time of pharmacokinetic analysis.
- Subject with lack of any measurable concentrations or only very low plasma concentrations.

NOTE: This exclusion will be assessed at the time of pharmacokinetic analysis.

# 8.1.2.2. Part 3 Multiple-Dose Pharmacokinetic Analysis Population

Part 3 Multiple-Dose Pharmacokinetic Analysis Population will include all subjects enrolled in Part 3 of the study, who are expected to provide evaluable pharmacokinetic data for the givinostat multiple-dose administration (Day 13), without deviations affecting pharmacokinetic interpretation.

The following reasons justify the exclusion of the pharmacokinetic data of a subject from the Part 3 multiple-dose pharmacokinetic analysis population:

 Protocol violation considered to have a potentially relevant effect on the pharmacokinetic results of the study.

NOTE: These protocol violations will be reported in the Data Blind Review Process Minute (Annex 5), and their impact will be assessed at the time of pharmacokinetic analysis.

- Subject experienced vomiting or diarrhea.
  - NOTE: Subjects that experienced vomiting or diarrhoea during this study part ill be reported in the Data Blind Review Process Minute (Annex 5), and their exclusion will be assessed at the time of pharmacokinetic analysis.
- Subject with lack of any measurable concentrations or only very low plasma concentrations.
   NOTE: This exclusion will be assessed at the time of pharmacokinetic analysis.

### 9. DATA REVIEW / TRANSFORMATION

### 9.1. Data Management

Data handling will be conducted in accordance with the Clinical Data Management section of the CSP and the Data Management Plan developed specifically for this study.

# 9.2. Acceptance of Data

For each study part, TFLs may start being programmed prior to or during the course of the trial. However, the programming of analysis datasets and TFLs will only be concluded and quality-controlled after database soft lock. Only audited data released by the bioanalytical laboratory will be used for programming the final analysis datasets and TFLs.

### 9.3. Data Transformation (CDISC)

Before performing the statistical analysis, all data collected (multiple sources) will be integrated into a common repository, using SAS® version 9.4 or higher.

For standardization and submission purpose, all data will be transformed according to Clinical Data Interchange Standards Consortium (CDISC):

Statistical Analysis Plan

EudraCT No: 2021-005756-11

- Study Data Tabulation Model (SDTM) version 1.4 or higher.
- SDTM Implementation Guide (SDTMIG) version 3.2 or higher.
- The following analysis datasets will be generated (Analysis Data Model [ADaM] version 2.1 or higher; ADaM Implementation Guide [ADaMIG], version 1.2 or higher) to support the results and ease the programming activities during the statistical analysis:
  - Subject-Level Analysis Dataset (ADSL).
  - Analysis Data Pharmacokinetic Concentrations (ADPC).
  - Analysis Data Pharmacokinetic Parameters (ADPP).
  - Analysis Data Adverse Events (ADAE).
  - Analysis Data Vital Signs (ADVS).
  - Analysis Data Electrocardiogram Parameters (ADEG).
  - Analysis Data Laboratory Test Results (ADLB).

For the scope of this trial, considering the primary and secondary objectives, six (6) Basic Data Structure (BDS) domains will be generated: ADPC, ADPP, ADAE, ADVS, ADEG and ADLB. These six datasets plus ADSL will be updated for each part. These domains will support the descriptive statistical analyses of the pharmacokinetic concentrations, the pharmacokinetic parameters and safety.

# ADSL - Subject-Level Analysis Dataset

This analysis domain will contain: general data about the subjects (i.e., age, sex and race), planned and actual allocated treatment analysis, and start and end dates of treatment analysis period. The origin of these data will primarily be the Demographics (DM) and Exposure (EX) SDTM domains. Besides this information, the following variables will be derived:

- Pharmacokinetic Analysis Set Population Flag 3 Subjects included in the Part 3 Single-Dose Pharmacokinetic Analysis Population.
- Pharmacokinetic Analysis Set Population Flag 4 Subjects included in the Part 3 Multiple-Dose Pharmacokinetic Analysis Population.
- Completers Population Flag Subjects who completed the treatment period.

# ADPC - Analysis Data Pharmacokinetic Concentrations

This is a BDS dataset that will contain the concentrations for each subject, per treatment analysis, per analyte/metabolite, and per timepoint.

The origin of these data will primarily be the EX and Pharmacokinetic Concentrations (PC) SDTM domains and ADSL ADaM domain.

Besides this information, the following variables will be derived:

- Pharmacokinetic Analysis Set Population Flag 1.
- Drug-Drug Interaction Analysis Set Population Flag 1
- Drug-Drug Interaction Analysis Set Population Flag 2
- Drug-Drug Interaction Analysis Set Population Flag 3.
- Drug-Drug Interaction Analysis Set Population Flag 4.
- Drug-Drug Interaction Analysis Set Population Flag 5.
- Drug-Drug Interaction Analysis Set Population Flag 6.
- Pharmacokinetic Analysis Set Population Flag 2.
- Drug-Drug Interaction Analysis Set Population Flag 7.
- Pharmacokinetic Analysis Set Population Flag 3.
- Pharmacokinetic Analysis Set Population Flag 4.

# ADPP - Analysis Data Pharmacokinetic Parameters

This is a BDS dataset that will contain the NCA pharmacokinetic parameters (plasma and urine) for each subject, per treatment analysis and per analyte/metabolite.

Besides the original pharmacokinetic parameter value, the dataset will contain the *ln*-transformed value that is necessary to apply for the specified statistical model(s).

The origin of these data will primarily be the DM and Pharmacokinetic Parameters (PP) SDTM domains.

Besides this information, the following variables will be derived:

- Pharmacokinetic Analysis Set Population Flag 1.
- Drug-Drug Interaction Analysis Set Population Flag 1.
- Drug-Drug Interaction Analysis Set Population Flag 2.
- Drug-Drug Interaction Analysis Set Population Flag 3.
- Drug-Drug Interaction Analysis Set Population Flag 4.
- Drug-Drug Interaction Analysis Set Population Flag 5.
- Drug-Drug Interaction Analysis Set Population Flag 6.
- Pharmacokinetic Analysis Set Population Flag 2.
- Drug-Drug Interaction Analysis Set Population Flag 7.
- Pharmacokinetic Analysis Set Population Flag 3.
- Pharmacokinetic Analysis Set Population Flag 4.

### ADAE - Analysis Data Adverse Events Dataset

This is an OCCDS dataset that will contain the adverse events for each subject.

The origin of these data will primarily be the Adverse Events (AE) SDTM domain and ADSL ADaM domain.

### ADVS - Analysis Data Vital Signs Dataset

This is a BDS dataset that will contain the vital signs results for each subject, per treatment analysis and per timepoint.

The origin of these data will primarily be the Vital Signs (VS) SDTM domain and ADSL ADaM domain.

### ADEG - Analysis Data Electrocardiogram Parameters Dataset

This is a BDS dataset that will contain the electrocardiogram for each subject, per treatment analysis and per timepoint.

The origin of these data will primarily be the ECG Test Results (EG) SDTM domain and ADSL ADaM domain.

# ADLB - Analysis Data Laboratory Test Results Dataset

This is a BDS dataset that will contain the safety laboratory test results for each subject and per treatment analysis.

The origin of these data will primarily be the Laboratory Test Results (LB) SDTM domain and ADSL ADaM domain.

### 10. STATISTICAL METHODS

### 10.1. General Considerations

Estimation of the pharmacokinetic parameters and drug-drug interaction comparative bioavailability analysis will be conducted on Phoenix<sup>®</sup> WinNonlin<sup>®</sup> version 8.2 or higher (Certara USA Inc, Princeton, NJ). All other statistical analysis will be conducted on SAS<sup>®</sup> version 9.4 or higher.

Statistical analyses and pharmacokinetic analyses will be performed in accordance with the U.S. FDA guidances [2, 3] and PPD applicable Standard Operating Procedures (SOPs).

Unless specified otherwise, continuous variables will be summarized with the following descriptive statistics: number of observations (n), mean, standard deviation (SD), minimum, median and maximum values. Categorical data will be summarized with frequencies and percentages. For subjects' characteristics and safety analyses, missing data will not be replaced; descriptive statistics and statistical analysis will be performed based on the available data only. All data recorded on discontinued subjects will be listed.

# 10.2. Subjects' Disposition

The number of subjects who completed each study part as well as subjects who withdrew prematurely from the study will be summarized by completion status and reason for withdrawal. Subjects who prematurely withdrew from the study will be listed.

The number of subjects included in each analysis population will be summarized, for each study part.

### 10.3. Protocol Deviations

During the respective Data Blind Review Process, all protocol deviations that occurred during each study part will be assessed in terms of their potential impact on the pharmacokinetic analysis. The result of this assessment will be reported in the respective Data Blind Review Process Minute (Annex 1, Annex 3, and Annex 5).

### 10.4. Plasma Pharmacokinetic Concentrations

For each study part (Part 1, Part 2 and Part 3), for the subjects included in the respective pharmacokinetic analysis population, descriptive statistics [n, geometric mean (G<sub>mean</sub>), arithmetic mean (A<sub>mean</sub>), SD, geometric SD (GSD), coefficient of variation (CV%), geometric CV% (GCV%), two-sided 95% CI of the A<sub>mean</sub> and G<sub>mean</sub>, median, minimum and maximum] of the plasma concentrations will be presented for each time point, by analyte, and by administration day. Concentrations below the LLOQ will be taken as missing for the calculation of the log-transformed statistics and as zero for the calculation of the remaining summary statistics.

Additionally, for Part 3, for the subjects included in the respective pharmacokinetic analysis population, descriptive statistics of the concentrations of givinostat and its metabolites in plasma will be presented by single and multiple-dose, and by sex.

Achievement of steady-state conditions will be determined by visual inspection of the trough plasma concentration-time profile (Ctrough). Analysis of variance of the plasma Ctrough may be performed if considered appropriate.

For each study part (Part 1, Part 2 and Part 3), individual (per subject) and G<sub>mess</sub> (including 95% CIs) plasma concentration versus time profile will be graphically displayed in both linear and semi-logarithmic scales:

- For plotting individual data in linear scale, concentrations below the LLOQ will be substituted by zero.
- For plotting G<sub>mean</sub> data in linear scale, concentrations below the LLOQ will be substituted by missing.
- For plotting data in semi-logarithmic scale, concentrations below the LLOQ before t<sub>max</sub>, will be substituted by ½ of the LLOQ value. After t<sub>max</sub>, concentrations below the LLOQ will be considered as missing. However, in case of two or more consecutive concentrations below the LLOQ, the first value will be replaced by ½ of the LLOQ value and the next values will be considered as missing.

Graphic presentation of individual data will be based on actual blood sampling time, except for predose sampling time which will be assumed as t<sub>0</sub>.

Concentration data from non-evaluable periods will be listed and graphically represented separately.

### 10.5. Plasma Pharmacokinetic Parameters

For each study part, plasma pharmacokinetic parameters will be calculated for the respective pharmacokinetic analysis population.

For each study part, for the subjects included in the pharmacokinetic analysis population, individual plasma pharmacokinetic parameters and descriptive statistics (n, G<sub>mean</sub>, A<sub>mean</sub>, SD, GSD, CV%, GCV%, two-sided 95% CI of the A<sub>mean</sub> and G<sub>mean</sub>, median, minimum and maximum), will be presented by investigational product.

If a given pharmacokinetic parameter could not be reliably determined for more than ½ of the subjects, only the minimum and maximum values will be presented, and the other descriptive statistics will be omitted for that parameter.

Missing pharmacokinetic parameter data will not be imputed.

For Part 3, for the subjects included in the respective pharmacokinetic analysis population, descriptive statistics of the plasma pharmacokinetic parameters of givinostat and its metabolites will be presented by single and multiple-dose, and by sex.

For Part 3, time dependency will be explored by comparing  $AUC_{0-\tau,ss}$  derived from the last dosing day (Day 13), after multiple doses administration, with  $AUC_{0-\infty}$  derived from the first dosing day (Day 1), after a single dose administration. Assessment of linearity will consider whether differences in AUC meet a criterion of  $\pm 25\%$ .

For Part 3, the Accumulation Index for  $C_{max}$  will be derived as the ratio  $\frac{C_{max,ss}}{C_{max}}$  and for AUC it will be derived as the ratio  $\frac{AUC_{0-T,ss}}{AUC_{0-t}}$ . Accumulation Index estimates will be summarized using  $A_{mean}$ , SD, SE median, minimum and maximum.

For Part 3, metabolic ratios will be calculated for each metabolite as 100 ·

ITF/2357/55 Version: 1.0 Date: 24MAR2022



 $\frac{AUC_{0-\infty,Metabolie}/MW_{Metabolite}}{AUC_{0-\infty,Givinostat}/MW_{Givinostat}}$ , for Day 1 (single-dose), and as 100  $\cdot \frac{AUC_{0-\tau,Metabolie}/MW_{Metabolite}}{AUC_{0-\tau,Givinostat}/MW_{Givinostat}}$ , for Day 13 (multiple-dose).

Note: MW represents the molecular weight of the analyte. For givinostat, MW is 421.49 g/mol; for ITF2374, MW is 405.49 g/mol; for ITF2375, MW is 406.47 g/mol; for ITF2440, MW is 257.33 g/mol; and for ITF2563, MW is 178.19 g/mol.

# 10.6. Urinary Data

For Part 3, for the subjects included in the pharmacokinetic analysis population, descriptive statistics (n, G<sub>mean</sub>, A<sub>mean</sub>, SD, GSD, CV%, GCV%, two-sided 95% CI of the A<sub>mean</sub> and G<sub>mean</sub>, median, minimum and maximum) of the urinary excretion profile and urinary cumulative excretion profile will be presented for each collection interval, by analyte, by single (Day 1) and multiple (Day 13) dose, and by sex. Concentrations below the LLOQ will be taken as missing for the calculation of the log-transformed statistics and as zero for the calculation of the remaining summary statistics.

Individual (per subject) and G<sub>mean</sub> urinary excretion versus time profile and urinary cumulative excretion versus time profile will be graphically displayed, in both linear and semi-logarithmic scales:

- For plotting individual data in linear scale, amounts below the LLOQ will be substituted by zero
- For plotting G<sub>mean</sub> data in linear scale, amounts below the LLOQ will be substituted by missing.

Day -1 sampling will be assumed as to.

### 10.7. Urinary Pharmacokinetic Parameters

For Part 3, urinary pharmacokinetic parameters will be calculated for the respective pharmacokinetic analysis population.

For Part 3, for the subjects included in the pharmacokinetic analysis population, individual urinary pharmacokinetic parameters and descriptive statistics (n, G<sub>mean</sub>, A<sub>mean</sub>, SD, GSD, CV%, GCV%, two-sided 95% CI of the A<sub>mean</sub> and G<sub>mean</sub>, median, minimum and maximum), will be presented by analyte, by single and multiple-dose, and by sex.

If a given pharmacokinetic parameter could not be reliably determined for more than \( \frac{1}{2} \) of the subjects, only the minimum and maximum values will be presented, and the other descriptive statistics will be omitted for that parameter.

Missing pharmacokinetic parameter data will not be imputed.

### 11. PRESENTATION OF RESULTS

### 11.1. Statistical Output Specification

Tables will be generated as Rich Text Files (\*.rtf) from SAS®.

Figures and Analysis Outputs will be generated as \*.docx files, exported from Phoenix WinNonlin®

and/or SAS®.

In-text Tables and Figures will preferably be prepared in portrait format. Listings will preferably be prepared in landscape format.

The CSR will be written according to PPD SOPs and templates for reporting bioavailability/bioequivalence trials.

# 11.2. Planned Tables, Figures, and Subject Data Listings

The planned Tables, Figures, and Individual Data Listings for the CSR are listed below.

# 11.2.1. In-text Tables and Figures

For CSR Synopsis:

The following Tables will be produced for direct insertion in the Synopsis of the CSR:

| Title |
|---|
| PART 3 |
| Givinostat and Its Main Metabolites (ITF2374 and ITF2375.): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Plasma |
| Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| Givinostat and Its Main Metabolites (ITF2374 and ITF2375,): Summary Statistics of the Plasma<br>Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Plasma |
| Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| Givinostat and Its Main Metabolites (ITF2374 and ITF2375): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Urinary |
| Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| Givinostat and Its Main Metabolites (ITF2374 and ITF2375): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Urinary |
| Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |

The following Figures will be produced for direct insertion in the Synopsis of the CSR:

| Legend |
|---|
| PART 3 |
| Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following |
| Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat. A - Linear |

| Legend | |
|---|---|
| Scale; B - Semi-I | ogarithmic Scale |
| <b>Profile Following</b> | olite (ITF2374): Geometric Mean (95% CI) Plasma Concentration Versus Time<br>Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of<br>). A – Linear Scale; B – Semi-Logarithmic Scale |
| <b>Profile Following</b> | blite (ITF2375): Geometric Mean (95% CI) Plasma Concentration Versus Time<br>Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of<br>). A – Linear Scale; B – Semi-Logarithmic Scale |
| <b>Profile Following</b> | blite (ITF2440): Geometric Mean (95% CI) Plasma Concentration <i>Versus</i> Time Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of ). A – Linear Scale; B – Semi-Logarithmic Scale |
| Givinostat Metabo<br>Profile Following | blite (ITF2563): Geometric Mean (95% CI) Plasma Concentration Versus Time<br>Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of<br>). A – Linear Scale; B – Semi-Logarithmic Scale |

# For CSR Body Text:

The following Tables and Figures will be produced for direct insertion in the body text of the CSR:

| In-text Tables | Title |
|---|---|
| PART 3 | |
| Table 3.A. | Study Flow-Chart – Part 3 |
| Table 3.B. | Identity of Investigational Products - Part 3 |
| Table 3.C. | Summary of Subjects Disposition – Part 3 |
| Table 3.D. | Summary of Demographic Data of the Pharmacokinetic Analysis Populations |
| Table 3.E. | Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563):<br>Summary Statistics of the Plasma Pharmacokinetic Parameters Following<br>Single-Dose Administration of Givinostat (Day 1) |
| Table 3.F. | Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563):<br>Summary Statistics of the Plasma Pharmacokinetic Parameters Following<br>Multiple-Dose Administration of Givinostat (Day 13) |
| Table 3.G. | Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563):<br>Summary Statistics of the Plasma Pharmacokinetic Parameters Accumulation<br>Index |
| Table 3.H. | Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563):<br>Summary Statistics of the Urinary Pharmacokinetic Parameters Following<br>Single-Dose Administration of Givinostat (Day 1) <sup>21</sup> |
| Table 3.I. | Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563):<br>Summary Statistics of the Urinary Pharmacokinetic Parameters Following<br>Multiple-Dose Administration of Givinostat (Day 13) <sup>21</sup> |
| Table 3.J. | Summary of Treatment-Emergent Adverse Events (TEAEs) |

| In-text Figures | Legend |
|---|---|
| PART 3 | |
| Figure 3.A.1. | Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time<br>Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13)<br>Administration of Givinostat – Linear Scale |
| Figure 3.A.2. | Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time<br>Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) |

| In-text Figures | Legend |
|---|---|
| | Administration of Givinostat - Semi-Logarithmic Scale |
| Figure 3.A.3. | Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time<br>Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day<br>13) – Linear Scale |
| Figure 3.A.4. | Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time<br>Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day<br>13) – Semi-Logarithmic Scale |
| Figure 3.A.5. | Givinostat: Geometric Mean (95% CI) Trough Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.B.1. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Single-Dose (Day 1) and<br>Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.B.2. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma<br>Concentration Versus Time Profile Following Single-Dose (Day 1) and<br>Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic<br>Scale |
| Figure 3.B.3. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.B.4. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma<br>Concentration Versus Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| Figure 3.B.5. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Trough Plasma<br>Concentration Versus Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.C.1. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Single-Dose (Day 1) and<br>Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.C.2. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma<br>Concentration Versus Time Profile Following Single-Dose (Day 1) and<br>Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic<br>Scale |
| Figure 3.C.3. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma<br>Concentration Versus Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.C.4. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| Figure 3.C.5. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Trough Plasma<br>Concentration Versus Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.D.1. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.D.2. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic |



| In-text Figures | Legend |
|---|---|
| | Scale |
| Figure 3.D.3. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration |
| | of Givinostat (Day 9 to Day 13) - Linear Scale |
| Figure 3.D.4. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| Figure 3.D.5. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Trough Plasma<br>Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.E.1. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Single-Dose (Day 1) and<br>Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.E.2. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma<br>Concentration Versus Time Profile Following Single-Dose (Day 1) and<br>Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic<br>Scale |
| Figure 3.E.3. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.E.4. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma<br>Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| Figure 3.E.5. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Trough Plasma<br>Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration<br>of Givinostat (Day 9 to Day 13) – Linear Scale |
| Figure 3.F.1. | Givinostat: Geometric Mean (95% CI) of Urinary Excretion Versus Time<br>Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13)<br>Administration of Givinostat – Linear Scale |
| Figure 3.F.2. | Givinostat: Geometric Mean (95% CI) of Cumulative Amount Urinary<br>Excretion <i>Versus</i> Time Profile Following Single-Dose (Day 1) and Multiple-<br>Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.G.1. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) of Urinary<br>Excretion <i>Versus</i> Time Profile Following Single-Dose (Day 1) and Multiple-<br>Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.G.2. | Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) of Cumulative<br>Amount Urinary Excretion <i>Versus</i> Time Profile Following Single-Dose (Day<br>1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.H.1. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) of Urinary<br>Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-<br>Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.H.2. | Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) of Cumulative<br>Amount Urinary Excretion <i>Versus</i> Time Profile Following Single-Dose (Day<br>1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.I.1. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) of Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.I.2. | Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) of Cumulative |

| In-text Figures | Legend |
|---|---|
| A | Amount Urinary Excretion Versus Time Profile Following Single-Dose (Day |
| | 1) and Multiple-Dose (Day 13) Administration of Givinostat - Linear Scale |
| Figure 3.J.1. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) of Urinary |
| | Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- |
| | Dose (Day 13) Administration of Givinostat - Linear Scale |
| Figure 3.J.2. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) of Cumulative |
| | Amount Urinary Excretion Versus Time Profile Following Single-Dose (Day |
| | 1) and Multiple-Dose (Day 13) Administration of Givinostat - Linear Scale |

# 11.2.2. Tables, Figures and Graphs Referred to But Not Included in the Text (Section 14 of CSR)

At least the following Tables and Figures should be produced for Section 14 of the CSR. If necessary, additional Tables and Figures should be prepared.

The following Tables and Figures will be compiled in a document, to be considered as Section 14 (Tables, Figures and Graph Referred To But Not Included in the Text) of the CSR.

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3. PART 3 | |
| 14.3.1. DEMOC | GRAPHIC DATA – PART 3 |
| 14.3.1.1. | Demographic Data – Part 3 Safety Analysis Population |
| 14.3.1.2. | Demographic Data – Part 3 Single-Dose Pharmacokinetic Analysis<br>Population |
| 14.3.1.3. | Demographic Data – Part 3 Multiple-Dose Pharmacokinetic Analysis<br>Population |
| 14.3.1.4. | Subjects Prematurely Discontinued After First Dosing |
| 14.3.2. PHARM | IACOKINETIC DATA – PART 3 |
| 14.3.2.1. | Plasma Pharmacokinetic Data |
| 14.3.2.1.1. | Deviations from Blood Sampling Schedule |
| 14.3.2.1.1.1. | Deviations from Blood Sampling Schedule |
| 14.3.2.1.1.2. | Missing Blood Samples |
| 14.3.2.1.1.3. | Other Important Protocol Deviations |
| 14.3.2.1.2. | Plasma Concentrations |
| 14.3.2.1.2.1. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Concentrations Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.2.2. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Concentrations Following Single-Dose Administration of Givinostat (Day 1)<br>– Male Subjects |
| 14.3.2.1.2.3. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Concentrations Following Single-Dose Administration of Givinostat (Day 1)<br>– Female Subjects |
| 14.3.2.1.2.4. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.1.2.5. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics<br>of Plasma Concentrations Following Single-Dose Administration of<br>Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.2.6. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.2.7. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.2.8. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics<br>of Plasma Concentrations Following Single-Dose Administration of<br>Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.2.9. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics<br>of Plasma Concentrations Following Single-Dose Administration of<br>Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.2.10. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.2.11. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.2.12. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.2.13. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.2.14. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.2.15. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics<br>of Plasma Concentrations Following Single-Dose Administration of<br>Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.2.16. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) |
| 14.3.2.1.2.17. | Givinostat: Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Male Subjects |
| 14.3.2.1.2.18. | Givinostat: Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Female Subjects |
| 14.3.2.1.2.19. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.1.2.20. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics<br>of Plasma Concentrations Following Multiple-Dose Administration of<br>Givinostat (Day 9 to Day 13) – Male Subjects |
| 14.3.2.1.2.21. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics<br>of Plasma Concentrations Following Multiple-Dose Administration of<br>Givinostat (Day 9 to Day 13) – Female Subjects |
| 14.3.2.1.2.22. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) |
| 14.3.2.1.2.23. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics<br>of Plasma Concentrations Following Multiple-Dose Administration of<br>Givinostat (Day 9 to Day 13) – Male Subjects |
| 14.3.2.1.2.24. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Female Subjects |
| 14.3.2.1.2.25. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) |
| 14.3.2.1.2.26. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Male Subjects |
| 14.3.2.1.2.27. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Female Subjects |
| 14.3.2.1.2.28. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) |
| 14.3.2.1.2.29. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Male Subjects |
| 14.3.2.1.2.30. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Female Subjects |
| 14.3.2.1.3. | Plasma Pharmacokinetic Parameters |
| 14.3.2.1.3.1. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Pharmacokinetic Parameters Following Single-Dose Administration of<br>Givinostat (Day 1) |
| 14.3.2.1.3.2. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Pharmacokinetic Parameters Following Single-Dose Administration of<br>Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.3.3. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Pharmacokinetic Parameters Following Single-Dose Administration of<br>Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.3.4. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.1.3.5. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.3.6. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.3.7. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.3.8. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.3.9. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.3.10. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.3.11. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.3.12. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.3.13. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.3.14. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.1.3.15. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.1.3.16. | Plasma Metabolic Ratios for Givinostat Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.3.17. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Pharmacokinetic Parameters Following Multiple-Dose Administration of<br>Givinostat (Day 13) |
| 14.3.2.1.3.18. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Pharmacokinetic Parameters Following Multiple-Dose Administration of<br>Givinostat ( Day 13) – Male Subjects |
| 14.3.2.1.3.19. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Pharmacokinetic Parameters Following Multiple-Dose Administration of<br>Givinostat (Day 13) – Female Subjects |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.1.3.20. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) |
| 14.3.2.1.3.21. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics |
| | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) - Male Subjects |
| 14.3.2.1.3.22. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics |
| | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.1.3.23. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics |
| | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) |
| 14.3.2.1.3.24. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics |
| | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) - Male Subjects |
| 14.3.2.1.3.25. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics |
| | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) - Female Subjects |
| 14.3.2.1.3.26. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics |
| | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) |
| 14.3.2.1.3.27. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics |
| | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) - Male Subjects |
| 14.3.2.1.3.28. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics |
| 3 | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) - Female Subjects |
| 14.3.2.1.3.29. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics |
| | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) |
| 14.3.2.1.3.30. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics |
| 11.5.2.1.5.50. | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.1.3.31. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics |
| 11.5.2.1.5.51. | of Plasma Pharmacokinetic Parameters Following Multiple-Dose |
| | Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.1.3.32. | Givinostat: Individual Data and Descriptive Statistics of Accumulation Index |
| 14.3.2.1.3.32. | Givinostat: Individual Data and Descriptive Statistics of Accumulation Index Givinostat: Individual Data and Descriptive Statistics of Accumulation Index |
| 14.5.2.1.5.55. | - Male Subjects |
| 14.3.2.1.3.34. | Givinostat: Individual Data and Descriptive Statistics of Accumulation Index |
| 11.5.2.1.5.51. | - Female Subjects |
| 14.3.2.1.3.35. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics |
| | of Accumulation Index |
| 14.3.2.1.3.36. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics |
| | of Accumulation Index – Male Subjects |
| 14.3.2.1.3.37. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics |
| 11.3.4.1.3.31. | of Accumulation Index – Female Subjects |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.1.3.38. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Accumulation Index |
| 14.3.2.1.3.39. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Accumulation Index – Male Subjects |
| 14.3.2.1.3.40. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Accumulation Index – Female Subjects |
| 14.3.2.1.3.41. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Accumulation Index |
| 14.3.2.1.3.42. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Accumulation Index – Male Subjects |
| 14.3.2.1.3.43. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Accumulation Index – Female Subjects |
| 14.3.2.1.3.44. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Accumulation Index |
| 14.3.2.1.3.45. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Accumulation Index – Male Subjects |
| 14.3.2.1.3.46. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Accumulation Index – Female Subjects |
| 14.3.2.1.3.47. | Plasma Metabolic Ratios for Givinostat Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.1.4. | Log-Linear Regression Parameters for λ <sub>z</sub> Estimation |
| 14.3.2.1.4.1. | Givinostat: Log-Linear Regression Parameters for λz Estimation Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.4.1. | Givinostat: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.4.2. | Givinostat Metabolite (ITF2374): Log-Linear Regression Parameters for λ <sub>z</sub><br>Estimation Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.4.3. | Givinostat Metabolite (ITF2375): Log-Linear Regression Parameters for λ <sub>z</sub><br>Estimation Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.4.4. | Givinostat Metabolite (ITF2440): Log-Linear Regression Parameters for λ <sub>z</sub><br>Estimation Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.4.5. | Givinostat Metabolite (ITF2563): Log-Linear Regression Parameters for $\lambda_z$<br>Estimation Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.4.6. | Givinostat: Log-Linear Regression Parameters for λ <sub>z</sub> Estimation Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.1.4.7. | Givinostat Metabolite (ITF2374): Log-Linear Regression Parameters for λ <sub>z</sub><br>Estimation Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.1.4.8. | Givinostat Metabolite (ITF2375): Log-Linear Regression Parameters for λ <sub>z</sub><br>Estimation Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.1.4.9. | Givinostat Metabolite (ITF2440): Log-Linear Regression Parameters for λ <sub>z</sub><br>Estimation Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.1.4.10. | Givinostat Metabolite (ITF2563): Log-Linear Regression Parameters for λ <sub>z</sub><br>Estimation Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2. | Urinary Pharmacokinetic Data |
| 14.3.2.2.1. | Deviations from Urine Sampling Schedule |
| 14.3.2.2.1.1. | Missing Urine Samples |


| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.2.2. | Urinary Excretion Profile |
| 14.3.2.2.2.1. | Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion<br>Profile Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.2.2. | Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion<br>Profile Following Single-Dose Administration of Givinostat (Day 1) – Male<br>Subjects |
| 14.3.2.2.2.3. | Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion<br>Profile Following Single-Dose Administration of Givinostat (Day 1) – Female<br>Subjects |
| 14.3.2.2.2.4. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.2.5. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.6. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.2.7. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.2.8. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.9. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.2.10. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.2.11. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.12. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.2.13. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.2.14. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.15. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics<br>of Urinary Excretion Profile Following Single-Dose Administration of<br>Givinostat (Day 1) – Female Subjects |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.2.2.16. | Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount<br>Urinary Excretion Profile Following Single-Dose Administration of<br>Givinostat (Day 1) |
| 14.3.2.2.2.17. | Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount<br>Urinary Excretion Profile Following Single-Dose Administration of<br>Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.18. | Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount<br>Urinary Excretion Profile Following Single-Dose Administration of<br>Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.2.19. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.2.20. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.1. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.2.22. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.2.3. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.24. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.25. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.2.26. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.7. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.2.8. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics<br>Cumulative Amount Urinary Excretion Profile Following Single-Dose<br>Administration of Givinostat (Day 1) |
| 14.3.2.2.2.29. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.2.30. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.2.31. | Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.2.2.32. | Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion<br>Profile Following Multiple-Dose Administration of Givinostat (Day 13) –<br>Male Subjects |
| 14.3.2.2.2.33. | Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion<br>Profile Following Multiple-Dose Administration of Givinostat (Day 13) –<br>Female Subjects |
| 14.3.2.2.2.34. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.2.35. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics<br>of Urinary Excretion Profile Following Multiple-Dose Administration of<br>Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.2.36. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.2.37. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.2.38. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics<br>of Urinary Excretion Profile Following Multiple-Dose Administration of<br>Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.2.39. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.2.40. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.2.41. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.2.42. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.2.43. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.2.44. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.2.45. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.2.46. | Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount<br>Urinary Excretion Profile Following Multiple-Dose Administration of<br>Givinostat (Day 13) |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.2.2.47. | Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount<br>Urinary Excretion Profile Following Multiple-Dose Administration of<br>Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.2.48. | Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount<br>Urinary Excretion Profile Following Multiple-Dose Administration of<br>Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.2.49. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.2.50. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.2.51. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.2.52. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.2.53. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.54. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.2.55. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.2.56. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.2.57. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.2.58. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics<br>Cumulative Amount Urinary Excretion Profile Following Multiple-Dose<br>Administration of Givinostat (Day 13) |
| 14.3.2.2.2.59. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.2.60. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.3. | Urinary Pharmacokinetic Parameters |
| 14.3.2.2.3.1. | Givinostat: Individual Data and Descriptive Statistics of Urinary<br>Pharmacokinetic Parameters Following Single-Dose Administration of<br>Givinostat (Day 1) |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.2.3.2. | Givinostat: Individual Data and Descriptive Statistics of Urinary<br>Pharmacokinetic Parameters Following Single-Dose Administration of<br>Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.3.3. | Givinostat: Individual Data and Descriptive Statistics of Urinary<br>Pharmacokinetic Parameters Following Single-Dose Administration of<br>Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.3.4. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.3.5. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.3.6. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.3.7. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.3.8. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.3.9. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.3.10. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.3.11. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.3.12. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.3.13. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.2.3.14. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects |
| 14.3.2.2.3.15. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects |
| 14.3.2.2.3.16. | Percentage of Dose Recovered in Urine for Givinostat and Givinostat<br>Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) Following Single-<br>Dose Administration of Givinostat (Day 1) |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.2.3.17. | Givinostat: Individual Data and Descriptive Statistics of Urinary<br>Pharmacokinetic Parameters Following Multiple-Dose Administration of<br>Givinostat (Day 13) |
| 14.3.2.2.3.18. | Givinostat: Individual Data and Descriptive Statistics of Urinary<br>Pharmacokinetic Parameters Following Multiple-Dose Administration of<br>Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.3.19. | Givinostat: Individual Data and Descriptive Statistics of Urinary<br>Pharmacokinetic Parameters Following Multiple-Dose Administration of<br>Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.3.20. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.3.21. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.3.22. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.3.23. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.3.24. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.3.25. | Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.3.26. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.3.27. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.3.28. | Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |
| 14.3.2.2.3.29. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| 14.3.2.2.3.30. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects |
| 14.3.2.2.3.31. | Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects |

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3.2.2.3.32. | Percentage of Dose Recovered in Urine for Givinostat and Givinostat Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) Following Multiple- |
| | Dose Administration of Givinostat (Day 13) |
| 14.3.3. SAFET | Y DATA – PART 3 |
| 14.3.3.1. | Adverse Events |
| 14.3.3.1.1. | Pre-Treatment Adverse Events |
| 14.3.3.1.2. | Treatment-Emergent Adverse Events (I) |
| 14.3.3.1.3. | Treatment-Emergent Adverse Events (II) |
| 14.3.3.2. | Vital Signs |
| 14.3.3.2.1. | Descriptive Statistics of Vital Signs Parameters |
| 14.3.3.2.2. | Descriptive Statistics of Change from Baseline of Vital Signs Parameters |
| 14.3.3.2.3. | Shifts in Vital Signs Parameters |
| 14.3.3.3. | 12-Lead ECG |
| 14.3.3.3.1. | Descriptive Statistics of 12-Lead ECG Parameters |
| 14.3.3.3.2. | Descriptive Statistics of Change from Baseline of 12-Lead ECG Parameters |
| 14.3.3.3.3. | Shifts in 12-Lead ECG Parameters |
| 14.3.3.4. | Hematology |
| 14.3.3.4.1. | Descriptive Statistics of Hematology Parameters |
| 14.3.3.4.2. | Descriptive Statistics of Change from Baseline of Hematology Parameters |
| 14.3.3.4.3. | Shifts in Hematology Parameters |
| 14.3.3.5. | Biochemistry |
| 14.3.3.5.1. | Descriptive Statistics of Biochemistry Parameters |
| 14.3.3.5.2. | Descriptive Statistics of Change from Baseline of Biochemistry Parameters |
| 14.3.3.5.3. | Shifts in Biochemistry Parameters |
| 14.3.3.6. | Coagulation |
| 14.3.3.6.1. | Descriptive Statistics of Coagulation Parameters |
| 14.3.3.6.2. | Descriptive Statistics of Change from Baseline of Coagulation Parameters |
| 14.3.3.6.3. | Shifts in Coagulation Parameters |
| 14.3.3.7. | Urinalysis |
| 14.3.3.7.1. | Descriptive Statistics of Urinalysis Parameters |
| 14.3.3.7.2. | Descriptive Statistics of Change from Baseline of Urinalysis Parameters |
| 14.3.3.7.3. | Shifts in Urinalysis Parameters |
| 14.3.3.8. | Body Weight |
| 14.3.3.8.1. | Descriptive Statistics of Body Weight |
| 14.3.3.8.2. | Descriptive Statistics of Body Weight - Male Subjects |
| 14.3.3.8.3. | Descriptive Statistics of Body Weight - Female Subjects |
| 14.3.3.8.4. | Descriptive Statistics of Change from Baseline of Body Weight |
| 14.3.3.8.5. | Descriptive Statistics of Change from Baseline of Body Weight – Male<br>Subjects |
| 14.3.3.8.6. | Descriptive Statistics of Change from Baseline of Body Weight – Female<br>Subjects |

| End-of-Text<br>Figures | Title |
|---|---|
| 14.3. PART 3 | |
| | ACOKINETIC DATA – PART 3 |
| 14.3.2.3. | Plasma Concentration Versus Time Profiles of All Subjects |
| 14.3.2.3.1. | Givinostat: Plasma Concentration Versus Time Profiles of All Subjects<br>Following Single-Dose Administration of Givinostat (Day 1) – Linear Scale |
| 14.3.2.3.2. | Givinostat: Plasma Concentration Versus Time Profiles of All Subjects<br>Following Multiple-Dose Administration of Givinostat (Day 13) – Linear<br>Scale |
| 14.3.2.3.3. | Givinostat Metabolite (ITF2374): Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) - Linear Scale |
| 14.3.2.3.4. | Givinostat Metabolite (ITF2374): Plasma Concentration <i>Versus</i> Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) – Linear Scale |
| 14.3.2.3.5. | Givinostat Metabolite (ITF2375): Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) - Linear Scale |
| 14.3.2.3.6. | Givinostat Metabolite (ITF2375): Plasma Concentration <i>Versus</i> Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) – Linear Scale |
| 14.3.2.3.7. | Givinostat Metabolite (ITF2440): Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) – Linear Scale |
| 14.3.2.3.8. | Givinostat Metabolite (ITF2440): Plasma Concentration <i>Versus</i> Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) – Linear Scale |
| 14.3.2.3.9. | Givinostat Metabolite (ITF2563): Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) - Linear Scale |
| 14.3.2.3.10. | Givinostat Metabolite (ITF2563): Plasma Concentration <i>Versus</i> Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) – Linear Scale |
| 14.3.2.4. | Individual Plasma Concentration Versus Time Profiles |
| 14.3.2.4.1. | Givinostat: Individual Plasma Concentration <i>Versus</i> Time Profile Following<br>Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of<br>Givinostat – Linear Scale |
| 14.3.2.4.2. | Givinostat: Individual Plasma Concentration Versus Time Profile Following<br>Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of<br>Givinostat – Semi-Logarithmic Scale |
| 14.3.2.4.3. | Givinostat: Individual Plasma Concentration <i>Versus</i> Time Profile Following<br>Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale |
| 14.3.2.4.4. | Givinostat: Individual Plasma Concentration <i>Versus</i> Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| 14.3.2.4.5. | Givinostat: Individual Trough Plasma Concentration Versus Time Profile<br>Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) –<br>Linear Scale |

| End-of-Text<br>Figures | Title |
|---|---|
| 14.3.2.4.6. | Givinostat Metabolite (ITF2374): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| 14.3.2.4.7. | Givinostat Metabolite (ITF2374): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale |
| 14.3.2.4.8. | Givinostat Metabolite (ITF2374): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale |
| 14.3.2.4.9. | Givinostat Metabolite (ITF2374): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| 14.3.2.4.10. | Givinostat Metabolite (ITF2374): Individual Trough Plasma Concentration<br>Versus Time Profile Following Multiple-Dose Administration of Givinostat<br>(Day 9 to Day 13) – Linear Scale |
| 14.3.2.4.11. | Givinostat Metabolite (ITF2375): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| 14.3.2.4.12. | Givinostat Metabolite (ITF2375): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale |
| 14.3.2.4.13. | Givinostat Metabolite (ITF2375): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale |
| 14.3.2.4.14. | Givinostat Metabolite (ITF2375): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| 14.3.2.4.15. | Givinostat Metabolite (ITF2375): Individual Trough Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale |
| 14.3.2.4.16. | Givinostat Metabolite (ITF2440): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| 14.3.2.4.17. | Givinostat Metabolite (ITF2440): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale |
| 14.3.2.4.18. | Givinostat Metabolite (ITF2440): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale |
| 14.3.2.4.19. | Givinostat Metabolite (ITF2440): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| 14.3.2.4.20. | Givinostat Metabolite (ITF2440): Individual Trough Plasma Concentration<br>Versus Time Profile Following Multiple-Dose Administration of Givinostat<br>(Day 9 to Day 13) – Linear Scale |



| End-of-Text<br>Figures | Title |
|---|---|
| 14.3.2.4.21. | Givinostat Metabolite (ITF2563): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| 14.3.2.4.22. | Givinostat Metabolite (ITF2563): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale |
| 14.3.2.4.23. | Givinostat Metabolite (ITF2563): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale |
| 14.3.2.4.24. | Givinostat Metabolite (ITF2563): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale |
| 14.3.2.4.25. | Givinostat Metabolite (ITF2563): Individual Trough Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale |
| 14.3.2.5. | Individual Urinary Excretion Versus Time Profiles |
| 14.3.2.5.1. | Givinostat: Individual Urinary Excretion Versus Time Profile Following<br>Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of<br>Givinostat – Linear Scale |
| 14.3.2.5.2. | Givinostat: Individual Cumulative Amount Urinary Excretion Versus Time<br>Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13)<br>Administration of Givinostat – Linear Scale |
| 14.3.2.5.3. | Givinostat Metabolite (ITF2374): Individual Urinary Excretion Versus Time<br>Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13)<br>Administration of Givinostat – Linear Scale |
| 14.3.2.5.4. | Givinostat Metabolite (ITF2374): Individual Cumulative Amount Urinary<br>Excretion <i>Versus</i> Time Profile Following Single-Dose (Day 1) and Multiple-<br>Dose (Day 13) Administration of Givinostat – Linear Scale |
| 14.3.2.5.5. | Givinostat Metabolite (ITF2375): Individual Urinary Excretion Versus Time<br>Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13)<br>Administration of Givinostat – Linear Scale |
| 14.3.2.5.6. | Givinostat Metabolite (ITF2375): Individual Cumulative Amount Urinary<br>Excretion <i>Versus</i> Time Profile Following Single-Dose (Day 1) and Multiple-<br>Dose (Day 13) Administration of Givinostat – Linear Scale |
| 14.3.2.5.7. | Givinostat Metabolite (ITF2440): Individual Urinary Excretion Versus Time<br>Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13)<br>Administration of Givinostat – Linear Scale |
| 14.3.2.5.8. | Givinostat Metabolite (ITF2440): Individual Cumulative Amount Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- Dose (Day 13) Administration of Givinostat – Linear Scale |
| 14.3.2.5.9. | Givinostat Metabolite (ITF2563): Individual Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| 14.3.2.5.10. | Givinostat Metabolite (ITF2563): Individual Cumulative Amount Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple- Dose (Day 13) Administration of Givinostat – Linear Scale |

# 11.2.3. List of Subject Data Listings (Section 16.2 of CSR)

The following Data Listings will be produced for Section 16.2. Subject Data Listings of the CSR.

If necessary, additional Data Listings should be prepared.

| Listing No. | Title |
|---|---|
| | TS DATA LISTING |
| 16.2.3. Part 3 | |
| 16.2.3.1. | Subject Disposition |
| 16.2.3.1.1. | Subject Disposition |
| 16.2.3.2. | Protocol Deviations |
| 16.2.3.2.1. | Blood Sampling Times Deviations |
| 16.2.3.2.2. | Other Protocol Deviations |
| 16.2.3.3. | Excluded Data from the Pharmacokinetic Analysis |
| 16.2.3.3.1. | Plasma Concentrations |
| 16.2.3.3.1.1. | Individual Data of Plasma Concentrations |
| 16.2.3.3.2. | Plasma Concentration Versus Time Profiles |
| 16.2.3.3.2.1. | Individual Plasma Concentration Versus Time Profiles - Linear Scale |
| 16.2.3.3.2.2. | Individual Plasma Concentration Versus Time Profiles – Semi-Logarithmic Scale |
| 16.2.3.3.3. | Urine Excretion |
| 16.2.3.3.3.1. | Individual Data of Plasma Concentrations |
| 16.2.3.3.4. | Urine Excretion Versus Time Profiles |
| 16.2.3.3.4.1. | Urine Excretion Versus Time Profiles – Linear Scale |
| 16.2.3.4. | Demographic and Other Baseline Data |
| 16.2.3.4.1. | Demographic Data |
| 16.2.3.4.2. | Fertility/Contraception |
| 16.2.3.4.2.1. | Female Fertility/Contraception |
| 16.2.3.4.2.2. | Male Fertility/Contraception |
| 16.2.3.4.3. | Drugs of Abuse, Ethanol and Cotinine |
| 16.2.3.4.4. | Viral Serology at Screening |
| 16.2.3.4.5. | Previous and Concomitant Medication |
| 16.2.3.4.6. | SARS-COV-2 Test |
| 16.2.3.5. | Compliance |
| 16.2.3.5.1. | Investigational Product Administration |
| 16.2.3.6. | Individual Pharmacokinetic Data |
| 16.2.3.6.1. | Givinostat: Individual Pharmacokinetic Data |
| 16.2.3.6.1.1. | Givinostat: Individual Drug Plasma Concentration Data |
| 16.2.3.6.1.2. | Givinostat: Individual Plasma Pharmacokinetic Parameters |
| 16.2.3.6.1.3. | Givinostat: Individual Plasma Pharmacokinetic Profiles |
| 16.2.3.6.1.4. | Givinostat: Individual Urine Excretion Data |
| 16.2.3.6.1.5. | Givinostat: Individual Urine Pharmacokinetic Parameters |
| 16.2.3.6.1.6. | Givinostat: Individual Urine Pharmacokinetic Profiles |
| 16.2.3.6.1.7. | Givinostat: Documentation of Statistical Analysis |
| 16.2.3.6.1.7.1. | Givinostat: Plasma Non-Compartmental Analysis Output |
| 16.2.3.6.1.7.2. | Givinostat: Plasma Non-Compartmental Analysis Plots |
| 16.2.3.6.1.7.3. | Givinostat: Urine Non-Compartmental Analysis Output |

| Listing No. | Title |
|---|---|
| 16.2.3.6.2. | Givinostat Metabolite (ITF2374): Individual Pharmacokinetic Data |
| 16.2.3.6.2.1. | Givinostat Metabolite (ITF2374): Individual Drug Plasma Concentration<br>Data |
| 16.2.3.6.2.2. | Givinostat Metabolite (ITF2374): Individual Plasma Pharmacokinetic<br>Parameters |
| 16.2.3.6.2.3. | Givinostat Metabolite (ITF2374): Individual Plasma Pharmacokinetic<br>Profiles |
| 16.2.3.6.2.4. | Givinostat Metabolite (ITF2374): Individual Urine Excretion Data |
| 16.2.3.6.2.5. | Givinostat Metabolite (ITF2374): Individual Urine Pharmacokinetic<br>Parameters |
| 16.2.3.6.2.6. | Givinostat Metabolite (ITF2374): Individual Urine Pharmacokinetic Profiles |
| 16.2.3.6.2.7. | Givinostat Metabolite (ITF2374): Documentation of Statistical Analysis |
| 16.2.3.6.2.7.1. | Givinostat Metabolite (ITF2374): Plasma Non-Compartmental Analysis<br>Output |
| 16.2.3.6.2.7.2. | Givinostat Metabolite (ITF2374): Plasma Non-Compartmental Analysis Plots |
| 16.2.3.6.2.7.3. | Givinostat Metabolite (ITF2374): Urine Non-Compartmental Analysis<br>Output |
| 16.2.3.6.3. | Givinostat Metabolite (ITF2375): Individual Pharmacokinetic Data |
| 16.2.3.6.3.1. | Givinostat Metabolite (ITF2375): Individual Drug Plasma Concentration<br>Data |
| 16.2.3.6.3.2. | Givinostat Metabolite (ITF2375): Individual Plasma Pharmacokinetic<br>Parameters |
| 16.2.3.6.3.3. | Givinostat Metabolite (ITF2375): Individual Plasma Pharmacokinetic<br>Profiles |
| 16.2.3.6.3.4. | Givinostat Metabolite (ITF2375): Individual Urine Excretion Data |
| 16.2.3.6.3.5. | Givinostat Metabolite (ITF2375): Individual Urine Pharmacokinetic<br>Parameters |
| 16.2.3.6.3.6. | Givinostat Metabolite (ITF2375): Individual Urine Pharmacokinetic Profiles |
| 16.2.3.6.3.7. | Givinostat Metabolite (ITF2375): Documentation of Statistical Analysis |
| 16.2.3.6.3.7.1. | Givinostat Metabolite (ITF2375): Plasma Non-Compartmental Analysis<br>Output |
| 16.2.3.6.3.7.2. | Givinostat Metabolite (ITF2375): Plasma Non-Compartmental Analysis Plot |
| 16.2.3.6.3.7.3. | Givinostat Metabolite (ITF2375): Urine Non-Compartmental Analysis<br>Output |
| 16.2.3.6.4. | Givinostat Metabolite (ITF2440): Individual Pharmacokinetic Data |
| 16.2.3.6.4.1. | Givinostat Metabolite (ITF2440): Individual Drug Plasma Concentration<br>Data |
| 16.2.3.6.4.2. | Givinostat Metabolite (ITF2440): Individual Plasma Pharmacokinetic<br>Parameters |
| 16.2.3.6.4.3. | Givinostat Metabolite (ITF2440): Individual Plasma Pharmacokinetic<br>Profiles |
| 16.2.3.6.4.4. | Givinostat Metabolite (ITF2440): Individual Urine Excretion Data |
| 16.2.3.6.4.5. | Givinostat Metabolite (ITF2440): Individual Urine Pharmacokinetic Parameters |
| 16.2.3.6.4.6. | Givinostat Metabolite (ITF2440): Individual Urine Pharmacokinetic Profiles |
| 16.2.3.6.4.7. | Givinostat Metabolite (ITF2440): Documentation of Statistical Analysis |
| 16.2.3.6.4.7.1. | Givinostat Metabolite (ITF2440): Plasma Non-Compartmental Analysis |

| Listing No. | Title |
|---|---|
| | Output |
| 16.2.3.6.4.7.2. | Givinostat Metabolite (ITF2440): Plasma Non-Compartmental Analysis Plots |
| 16.2.3.6.4.7.3. | Givinostat Metabolite (ITF2440): Urine Non-Compartmental Analysis<br>Output |
| 16.2.3.6.5. | Givinostat Metabolite (ITF2563): Individual Pharmacokinetic Data |
| 16.2.3.6.5.1. | Givinostat Metabolite (ITF2563): Individual Drug Plasma Concentration<br>Data |
| 16.2.3.6.5.2. | Givinostat Metabolite (ITF2563): Individual Plasma Pharmacokinetic<br>Parameters |
| 16.2.3.6.5.3. | Givinostat Metabolite (ITF2563): Individual Plasma Pharmacokinetic<br>Profiles |
| 16.2.3.6.5.4. | Givinostat Metabolite (ITF2563): Individual Urine Excretion Data |
| 16.2.3.6.5.5. | Givinostat Metabolite (ITF2563): Individual Urine Pharmacokinetic<br>Parameters |
| 16.2.3.6.5.6. | Givinostat Metabolite (ITF2563): Individual Urine Pharmacokinetic Profiles |
| 16.2.3.6.5.7. | Givinostat Metabolite (ITF2563): Documentation of Statistical Analysis |
| 16.2.3.6.5.7.1. | Givinostat Metabolite (ITF2563): Plasma Non-Compartmental Analysis<br>Output |
| 16.2.3.6.5.7.2. | Givinostat Metabolite (ITF2563): Plasma Non-Compartmental Analysis Plots |
| 16.2.3.6.5.7.3. | Givinostat Metabolite (ITF2563): Urine Non-Compartmental Analysis<br>Output |
| 16.2.3.7. | Adverse Event Listings (Each Subject) |
| 16.2.3.7.1. | Pre-Treatment Adverse Events |
| 16.2.3.7.2. | Treatment-Emergent Adverse Events |
| 16.2.3.7.3. | Serious Adverse Events (I) |
| 16.2.3.8. | Listings of Laboratory Measurements by Subject |
| 16.2.3.8.1. | Normal Range of Laboratory Values |
| 16.2.3.8.2. | Hematology (I) |
| 16.2.3.8.3. | Hematology (II) |
| 16.2.3.8.4. | Biochemistry (I) |
| 16.2.3.8.5. | Biochemistry (II) |
| 16.2.3.8.6. | Biochemistry (III) |
| 16.2.3.8.7. | Biochemistry (IV) |
| 16.2.3.8.8. | Biochemistry (V) |
| 16.2.3.8.9. | Coagulation |
| 16.2.3.8.10. | Urinalysis |
| 16.2.3.8.11. | Urine Microscopy |
| 16.2.3.8.12. | Pregnancy Test |
| 16.2.3.8.13. | Additional (Not Planned) Laboratory Safety Tests |
| 16.2.3.9. | Vital Signs |
| 16.2.3.10. | 12-Lead ECG |
| 16.2.3.11. | Urine Sampling |

Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 12. REFERENCES

- [1] ITF/2357/55 Clinical Study Protocol, Version 1.0, 29NOV2021
- [2] Food and Drug Administration (FDA), Clinical Drug Interaction Studies Cytochrome P450 Enzyme- and Transporter-Mediated Drug Interactions Guidance for Industry (2020).

# 13. APPENDICES

APPENDIX A. Planned Tables, Figures, and Subject Data Listings

A.1. In-text Tables and Figures - For CSR Synopsis

#### A.1.1. Part 3

#### SYNOPSIS TABLES (1)

Givinostat and Its Main Metabolites (ITF2374 and ITF2375,): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1)

| Parameter (unit) | Givinostat $(n = xx)$ | ITF2374<br>(n = xx) | ITF2375<br>(n = xx) |
|---|---|---|---|
| C <sub>max</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| T <sub>max</sub> (h) | xx.xx(xx.xx-xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx (xx.xx - xx.xx) |
| AUCot ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| AUC₀∞ ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| %AUCextrap (%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $\lambda_z(1/h)$ | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) |
| t <sub>1/2</sub> (h) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |

n - Number of Subjects

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n = xx, for < Investigational Product > product > product > roduct >

Values are geometric mean (Gmoun) with geometric coefficient of variation (GCV%) within parenthesis

T<sub>max</sub> values are median with range between parentheses

# SYNOPSIS TABLES (2)

Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1)

| Parameter (unit) | $ \begin{array}{c} \text{ITF2440} \\ \text{(n = xx)} \end{array} $ | $ \begin{array}{c} \text{ITF2563} \\ \text{(n = xx)} \end{array} $ |
|---|---|---|
| C <sub>max</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| T <sub>max</sub> (h) | xx.xx(xx.xx-xx.xx) | xx.xx(xx.xx - xx.xx) |
| AUC <sub>0-t</sub> ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| AUC₀∞ ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| %AUC <sub>extrap</sub> (%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $\lambda_z(1/h)$ | x.xxx (xx.x%) | x.xxx (xx.x%) |
| t <sub>16</sub> (h) | xx.xx (xx.x%) | xx.xx (xx.x%) |

n - Number of Subjects

Values are geometric mean (Gmosm) with geometric coefficient of variation (GCV%) within parenthesis

T<sub>max</sub> values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For <Parameter(s)>, n=xx, for <Investigational Product> product> and n=xx, for <Investigational Product> product>'.

# SYNOPSIS TABLES (3)

Givinostat and Its Main Metabolites (ITF2374 and ITF2375,): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13)

| Parameter (unit) | Givinostat<br>(n = xx) | ITF2374<br>(n = xx) | $ \begin{array}{l} \text{ITF 2375} \\ \text{(n = xx)} \end{array} $ |
|---|---|---|---|
| C <sub>max,ss</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| T <sub>max,55</sub> (h) | xx.xx(xx.xx-xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx (xx.xx - xx.xx) |
| AUC <sub>0-T,SS</sub> ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| AUC <sub>0-t</sub> ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| AUC₀∞ ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $\lambda_z (1/h)$ | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) |
| t <sub>1/2</sub> (h) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| CL <sub>ss</sub> /F (L/h) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| V <sub>D</sub> /F (L) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |

n - Number of Subjects

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > product > roduct > r

Values are geometric mean (Gmean) with geometric coefficient of variation (GCV%) within parenthesis

T<sub>max</sub> values are median with range between parentheses

# SYNOPSIS TABLES (4)

Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13)

| Parameter (unit) | $ \begin{array}{l} \text{ITF2440} \\ \text{(n = xx)} \end{array} $ | ITF2563<br>(n = xx) |
|---|---|---|
| C <sub>max,55</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| T <sub>max,55</sub> (h) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) |
| AUC <sub>0-t,ss</sub> ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| AUC <sub>0-t</sub> ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| AUC₀∞ ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| $\lambda_z(1/h)$ | x.xxx (xx.x%) | x.xxx (xx.x%) |
| t34 (h) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| CL <sub>ss</sub> /F (L/h) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| V <sub>D</sub> /F (L) | xx.xx (xx.x%) | xx.xx (xx.x%) |

n - Number of Subjects

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the #symbol and accompanied by a footnote: '# For <Parameter(s)>, n=xx, for <Investigational Product> product> '.

Values are geometric mean (Gmean) with geometric coefficient of variation (GCV%) within parenthesis

T<sub>max</sub> values are median with range between parentheses

# SYNOPSIS TABLES (5)

Givinostat and Its Main Metabolites (ITF2374 and ITF2375): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) 10

#### SYNOPSIS TABLES (6)

Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1)  $^{II}$ 

# SYNOPSIS TABLES (7)

Givinostat and Its Main Metabolites (ITF2374 and ITF2375): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 10

#### SYNOPSIS TABLES (8)

Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 11

10 To be generated as follows:

| Parameter (unit) | Givinostat $(n = xx)$ | $ ITF2374 \\ (n = xx) $ | ITF2375<br>(n = xx) |
|---|---|---|---|
| R <sub>max,55</sub> ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| tu <sub>max</sub> (h) | xx.xx(xx.xx - xx.xx) | xx.xx(xx.xx - xx.xx) | xx.xx (xx.xx - xx.xx) |
| Amt <sub>CUM</sub> ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| AURCo+ ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| REC% (%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| CL <sub>R</sub> /F (L/h) | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) |

n - Number of Subjects

Values are geometric mean (Gmean) with geometric coefficient of variation (GCV%) within parenthesis

tumax values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3
Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > product > roduct > r

11 To be generated as follows:

| Parameter (unit) | $ \begin{array}{l} \mathbf{ITF2440} \\ \mathbf{(n = xx)} \end{array} $ | ITF2563<br>(n = xx) |
|---|---|---|
| R <sub>max,ss</sub> ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| tu <sub>max</sub> (h) | xx.xx(xx.xx - xx.xx) | xx.xx (xx.xx - xx.xx) |
| Amt <sub>CUM</sub> ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| AURCo+ ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) |
| REC% (%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| CL <sub>R</sub> /F (L/h) | x.xxx (xx.x%) | x.xxx (xx.x%) |

n - Number of Subjects

Values are geometric mean (Gmosn) with geometric coefficient of variation (GCV%) within parenthesis tumax values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > roduct > ro

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# SYNOPSIS FIGURES (9)

Givinostat: Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat. A – Linear Scale; B – Semi-Logarithmic Scale

#### SYNOPSIS FIGURES (10)

Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat (Day 1). A – Linear Scale; B – Semi-Logarithmic Scale

#### SYNOPSIS FIGURES (11)

Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat (Day 1). A – Linear Scale; B – Semi-Logarithmic Scale

#### SYNOPSIS FIGURES (12)

Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat (Day 1). A – Linear Scale; B – Semi-Logarithmic Scale

#### SYNOPSIS FIGURES (13)

Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma Concentration *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat (Day 1). A – Linear Scale; B – Semi-Logarithmic Scale

# A.2. In-text Tables and Figures - For CSR Body Text

# A.2.1. Part 3

# Table 1.A. Study Flow-Chart - Part 3

Note: To be captured from the Clinical Study Protocol (CSP) and Amendments.

# Table 1.B. Identity of Investigational Products - Part 3

Note: To be generated by the Medical Writing (MW).

# Table 1.C. Summary of Subjects Disposition - Part 3

| Disposition | Number of<br>Subjects |
|--------------------------------------------|-----------------------|
| Admitted to Treatment Period | ZZ |
| Discontinued after First Dosing | 77 |
| Reason - < Reason > | xx |
| Part 3 Safety Analysis Population | XX |
| Part 3 Pharmacokinetic Analysis Population | XX |
| Completed Part 3 of Study | XX |

Program: <SAS Program>



Table 1.D. Summary of Demographic Data of the Pharmacokinetic Analysis Populations

| Demography | Parameter | Single-Dose | Multiple-Dose |
|-----------------------|------------------|-------------|---------------|
| Age (years) | n | xx | xx |
| | Mean | XX | xx |
| | SD | XX.X | XX,X |
| | Median | xx | xx |
| | Minimum | xx | XX |
| | Maximum | xx | XX |
| Sex, n (%) | n | XX | XX |
| | Male | xx (xx.x%) | xx (xx.x%) |
| | Female | xx (xx.x%) | xx (xx.x%) |
| Race, n (%) | n | xx | XX |
| | <race></race> | xx (xx.x%) | xx (xx.x%) |
| Weight (kg) | n | xx | XX |
| 7.00 | Mean | XX.X | XX.X |
| | SD | xx.xx | XX.XX |
| | Median | XX.X | XX.X |
| | Minimum | xx.x | XX.X |
| | Maximum | XX.X | XX.X |
| Height (cm) | n | XX | XX |
| 4.2010 p | Mean | xxx | XXX |
| | SD | XX.X | XX.X |
| | Median | xxx | XXX |
| | Minimum | xxx | XXX |
| | Maximum | xxx | xxx |
| Body Mass Index (kg/m | <sup>2</sup> ) n | xx | XX |
| | Mean | XX.X | XX.X |
| | SD | xx.xx | xx.xx |
| | Median | xx.x | XX.X |
| | Minimum | XX.X | XX.X |
| | Maximum | xx.x | XX.X |

n - Number of Subjects; SD - Standard Deviation

Program: <SAS Program>

Table 1.E. Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1)

| | | $(\mathbf{n} = \mathbf{x}\mathbf{x})$ | $(\mathbf{n} = \mathbf{x}\mathbf{x})$ | $(\mathbf{n} = \mathbf{x}\mathbf{x})$ |
|---|---|---|---|---|
| xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| xx.xx - xx.xx | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| xx.xx (xx.xx –<br>xx.xx) | xx.xx (xx.xx -<br>xx.xx) | xx.xx (xx.xx -<br>xx.xx) | xx.xx (xx.xx –<br>xx.xx) | xx.xx (xx.xx -<br>xx.xx) |
| xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| xx.xx - xx.xx | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| 2 7 7 7 7 | xx.xx (xx.xx - xx.xx)<br>xx.xx (xx.x%)<br>xx.xx - xx.xx]<br>xx.xx - xx.xx]<br>xx.xx - xx.xx]<br>xx.xx - xx.xx]<br>xx.xx (xx.x%)<br>xx.xx - xx.xx]<br>xx.xx (xx.x%) | XX.XX (XX.XX - XX.XX (XX.XX - XX.XX) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX - XX.XX XX.XX (XX.X%) XX.XX - XX.XX [XX.XX - XX.XX] XX.XX (XX.X%) XX.XX (XX.X%) XX.XX - XX.XX [XX.XX - XX.XX] XX.XX (XX.X%) XX.XX (XX.X%) XX.XX - XX.XX [XX.XX - XX.XX] XX.XX - XX.XX [XX.XX - XX.XX] XX.XX (XX.X%) XX.XX (XX.X%) | XX.XX (XX.XX - XX.XX (XX.XX - XX.XX) XX.XX) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) | XX.XX (XX.XX - XX.XX (XX.XX - XX.XX) XX.XX) XX.XX) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] [XX.XX - XX.XX] XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) XX.XX (XX.X%) |

n - Number of Subjects

Values are geometric mean (G<sub>mean</sub>) with geometric coefficient of variation (GCV%) within parenthesis and 95% confidence interval of the G<sub>mean</sub> within square brackets

T<sub>max</sub> values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > product > roduct > r

Table 1.F. Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13)

| Parameter (unit) | Givinostat<br>(n = xx) | ITF2374<br>(n = xx) | ITF2375<br>(n = xx) | ITF2440<br>(n = xx) | ITF2563<br>(n = xx) |
|---|---|---|---|---|---|
| C <sub>max,ss</sub> ( <unitsc>)</unitsc> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| T <sub>max,ss</sub> (h) | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | (xx.xx - xx.xx) | (xx.xx - xx.xx) | (xx.xx - xx.xx) | (xx.xx - xx.xx) | (xx.xx - xx.xx) |
| AUC <sub>0-t,ss</sub> ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| AUC <sub>0-t</sub> ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| CALLES CO. | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| AUC₀∞ ( <unitsa>)</unitsa> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| $\lambda_z (1/h)$ | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) | x.xxx (xx.x%) |
| 2.40.0 | [x.xxx - x.xxx] | [x.xxx - x.xxx] | [x.xxx - x.xxx] | [x.xxx - x.xxx] | [x.xxx - x.xxx] |
| t <sub>1/2</sub> (h) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| CL <sub>ss</sub> /F (L/h) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| V <sub>D</sub> /F (L) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| 3.0 | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |

n - Number of Subjects

Values are geometric mean (Gmoan) with geometric coefficient of variation (GCV%) within parenthesis and 95% confidence interval of the Gmoan within square brackets

Tmax,ss values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the #symbol and accompanied by a footnote: '#For <Parameter(s)>, n=xx, for <Investigational Product> product> '.

# Table 1.G. Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563): Summary Statistics of the Plasma Pharmacokinetic Parameters Accumulation Index

| Parameter (unit) | Givinostat<br>(n = xx) | ITF2374<br>(n = xx) | ITF2375<br>(n = xx) | ITF2440<br>(n = xx) | ITF2563<br>(n = xx) |
|---|---|---|---|---|---|
| C <sub>max</sub> | xx.xx ± xx.xx | xx.xx ± xx.xx | xx.xx ± xx.xx | xx.xx ± xx.xx | xx.xx ± xx.xx |
| C <sub>max</sub><br>AUC <sub>0-t</sub> | $xx.xx \pm xx.xx$ | $xx.xx \pm xx.xx$ | $xx.xx \pm xx.xx$ | $xx.xx \pm xx.xx$ | $xx.xx \pm xx.xx$ |

n - Number of Subjects

Values are arithmetic mean (Amean) ± standard deviation

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3 Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the #symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product >, and n=xx, for < Investigational Product > product >'.

Table 1.H. Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) 21

Table 1.I. Givinostat and Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 21

### 1 To be generated as follows:

| Parameter (unit) | Givinostat<br>(n = xx) | ITF2374<br>(n = xx) | ITF2375<br>(n = xx) | $ \text{ITF2440} \\ (n = xx) $ | ITF2563<br>(n = xx) |
|---|---|---|---|---|---|
| R <sub>max,55</sub> ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| tu <sub>max</sub> (h) | xx.xx (xx.xx -<br>xx.xx) | xx.xx (xx.xx -<br>xx.xx) | xx.xx (xx.xx -<br>xx.xx) | xx.xx (xx.xx -<br>xx.xx) | xx.xx (xx.xx -<br>xx.xx) |
| Amtcum ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| O STATE OF THE PARTY OF THE PAR | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| AURCo+ ( <units>)</units> | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| REC% (%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |
| CL <sub>R</sub> /F (L/h) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) | xx.xx (xx.x%) |
| | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] | [xx.xx - xx.xx] |

n - Number of Subjects

Values are geometric mean ( $G_{mean}$ ) with geometric coefficient of variation (GCV%) within parenthesis and 95% confidence interval of the  $G_{mean}$  within square brackets

tumax values are median with range between parentheses

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: This table will present the summary statistics of the pharmacokinetic parameters calculated for Part 3
Pharmacokinetic Analysis Population. In case a pharmacokinetic parameter could not be calculated for one or more subjects in the Part 1 Pharmacokinetic Analysis Population, the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > product > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) >, n=xx, for < Investigational Product > product > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter(s) > content of the pharmacokinetic parameter should be followed by the # symbol and accompanied by a footnote: '# For < Parameter should be followed by the # symbol and accompanied by a footnote should be followed by the # symbol and accompanied by the # symbol and accompanied by the # symbol and accompanied by the # symbol and accompanied by



Table 1.J. Summary of Treatment-Emergent Adverse Events (TEAEs)

| | Total (N = xx) | |
|---|---|---|
| | All TEAEs | Drug-related TEAEs |
| Number of Subjects {Nr. of<br>TEAEs} (% of Subjects) | xx {xx} (xx%) | xx {xx} (xx%) |
| MedDRA | | |
| System Organ Class (SOC)<br>Preferred Term (PT) | | |
| <teaes soc=""></teaes> | xx {xx} (xx%) | xx {xx} (xx%) |
| <teaes soc=""></teaes> | xx {xx} (xx%) | xx {xx} (xx%) |
| Sinsert as many rows as deemed necessary | | |
| Severity | | |
| Mild | xx {xx} (xx%) | xx {xx} (xx%) |
| Moderate | xx {xx} (xx%) | xx {xx} (xx%) |
| Severe | xx {xx} (xx%) | xx {xx} (xx%) |

MedDRA - Medical Dictionary for Regulatory Activities

Drug-related TEAEs are those which causality was assessed as "Reasonably Possible" by the Investigator.

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- Figure 1.A.1. Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- Figure 1.A.2. Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Semi-Logarithmic Scale
- Figure 1.A.3. Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale
- Figure 1.A.4. Givinostat: Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Semi-Logarithmic Scale
- Figure 1.A.5. Givinostat: Geometric Mean (95% CI) Trough Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale
- Figure 1.B.1. Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale
- Figure 1.B.2. Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale
- Figure 1.B.3. Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale
- Figure 1.B.4. Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale
- Figure 1.B.5. Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) Trough Plasma Concentration *Versus* Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale



- Figure 1.C.1. Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale
- Figure 1.C.2. Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale
- Figure 1.C.3. Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale
- Figure 1.C.4. Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale
- Figure 1.C.5. Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) Trough Plasma Concentration *Versus* Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale
- Figure 1.D.1. Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale
- Figure 1.D.2. Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale
- Figure 1.D.3. Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale
- Figure 1.D.4. Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale
- Figure 1.D.5. Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) Trough Plasma Concentration *Versus* Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- Figure 1.E.1. Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale
- Figure 1.E.2. Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale
- Figure 1.E.3. Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale
- Figure 1.E.4. Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Semi-Logarithmic Scale
- Figure 1.E.5. Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) Trough Plasma Concentration *Versus* Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

Figure 1.F.1. Givinostat: Geometric Mean (95% CI) of Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.F.2. Givinostat: Geometric Mean (95% CI) of Cumulative Amount Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.G.1. Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) of Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.G.2. Givinostat Metabolite (ITF2374): Geometric Mean (95% CI) of Cumulative Amount Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.H.1. Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) of Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.H.2. Givinostat Metabolite (ITF2375): Geometric Mean (95% CI) of Cumulative Amount Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.I.1. Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) of Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.I.2. Givinostat Metabolite (ITF2440): Geometric Mean (95% CI) of Cumulative Amount Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.J.1. Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) of Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Figure 1.J.2. Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) of Cumulative Amount Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# A.3. Tables, Figures and Graphs Referred to But Not Included in the Text (Section 14 of CSR)

#### 14.1.1. SAFETY DATA -

A.3.1. Part 3

#### 14.2. PART 3

#### 14.2.1. DEMOGRAPHIC DATA - PART 3

14.2.1.1. Demographic Data - Part 3 Safety Analysis Population 2

14.2.1.2. Demographic Data - Part 3 Single-Dose Pharmacokinetic Analysis Population 2

14.2.1.3. Demographic Data – Part 3 Multiple-Dose Pharmacokinetic Analysis Population 2

<sup>2</sup> To be generated as follows:

| Subject No. | Sex | Race | Age<br>(years) | Height (cm) | Weight<br>(kg) | BMI<br>(kg/m²) |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | <male <br="">Female&gt;</male> | <race></race> | xx | xxx | XX.X | XX.X |
| <insert as="" man<="" td=""><td>y rows as deer</td><td>ned necessary&gt;</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td></insert> | y rows as deer | ned necessary> | XX | XX | XX | XX |
| | | Mean | XX | XXX | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.XX | XX XX |
| | | Median | XX | XXX | XX.X | XX.X |
| | | Minimum | XX | XXX | XX.X | XX.X |
| | | Maximum | XX | XXX | XX.X | XX.X |

BMI - Body Mass Index; n - Number of Subjects; SD - Standard Deviation

Program: <SAS Program>

Execution Date/Time: <a href="mailto:sddMMMyyyyHH:MM">ddMMMyyyy HH:MM</a>

#### 14.2.1.4. Subjects Prematurely Discontinued After First Dosing

| Subject No. | Time of Discontinuation | Reason for Discontinuation |
|---|---|---|
| <subject id=""> <day #=""></day></subject> | | <reason></reason> |
| <insert as="" many="" rows<="" td=""><td>as deemed necessary&gt;</td><td></td></insert> | as deemed necessary> | |

Program: <SAS Program>

### 14.2.2. PHARMACOKINETIC DATA - PART 3

#### 14.2.2.1. Plasma Pharmacokinetic Data

# 14.2.2.1.1. Deviations from Blood Sampling Schedule

# 14.2.2.1.1.1. Deviations from Blood Sampling Schedule

| Subject No. | Day of<br>Dose | Analyte | Planned<br>Time<br>(h:min) | Deviation (h:min) Reason for Deviation |
|---|---|---|---|---|
| <subject></subject> | <day #=""></day> | <analyte></analyte> | <planned<br>blood<br/>sampling<br/>time&gt;</planned<br> | <deviation<reason (e.g.="" blood="" deviation="" difficulty="" for="" time="" with=""> sampling / Subject unavailable at scheduled time)&gt;</deviation<reason> |

<Insert as many rows as deemed necessary>

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

# 14.2.2.1.1.2. Missing Blood Samples

| Subject No. | Day of<br>Dose | Analyte | Planned Time<br>(h:min) | Reason for Missing Blood Sample |
|---|---|---|---|---|
| <subject id=""></subject> | <day#></day#> | <analyte></analyte> | <planned blood="" sampling="" time=""></planned> | <reason blood="" for="" missing="" sample=""></reason> |
| <insert as<br="">many rows as<br/>deemed<br/>necessary&gt;</insert> | | | | |

Program: <SAS Program>
Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 14.2.2.1.1.3. Other Important Protocol Deviations

| Subject No. | Day of Dose | Analyte | Category | Description |
|---|---|---|---|---|
| <subject id=""></subject> | <day #=""></day> | <analyte></analyte> | <deviation category=""></deviation> | <description deviation="" of=""></description> |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | |

Program: <SAS Program>

Execution Date/Time: <a href="mailto:</a><a href="mailto:ddMMMyyyy HH:MM">ddMMMyyyy HH:MM</a></a>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### 14.2.2.1.2. Plasma Concentrations

- 14.2.2.1.2.1. Givinostat: Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1)  $^3$
- 14.2.2.1.2.2. Givinostat: Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.2.3. Givinostat: Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.1.2.4. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.1.2.5. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.2.6. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.1.2.7. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) <sup>3</sup>
- 14.2.2.1.2.8. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.2.9. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.1.2.10. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.1.2.11. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.2.12. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Female Subjects  $^3$
- 14.2.2.1.2.13. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.1.2.14. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.2.15. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>

Date: <DDMMMYYYY>

<sup>3</sup> To be generated as follows:

| To be generaled as jollows. | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject No. | Pre-dose - | | | | | Time Pos | st-Dose (h) | | | | |
| Subject No. | 11e-dose | X.XX | Z.XX | X.XX | Z.XX | X.XX | ZZ.Z | 7.77 | X.XX | X.XX | 7.77 |
| <subject id=""></subject> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| <insert as="" deemed="" many="" r<="" rows="" td=""><td>necessary&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></insert> | necessary> | | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Gmean ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GSD ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Gmean 95% CI Upper ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean 95% CI Lower ( units C ) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean 95% CI Upper ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

n – Number of Subjects; Gmean – Geometric Mean; Amean – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

BLQ - Below the Limit of Quantification (LLOQ = <LLOQ> <unitsC>) of the assay (taken as missing for the calculation of log-transformed statistics and as zero for the calculation of the remaining summary statistics)

ND - Not Done

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- 14.2.2.1.2.16. Givinostat: Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) 4
- 14.2.2.1.2.17. Givinostat: Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Male Subjects <sup>4</sup>
- 14.2.2.1.2.18. Givinostat: Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Female Subjects 4
- 14.2.2.1.2.19. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) 4
- 14.2.2.1.2.20. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Male Subjects <sup>4</sup>
- 14.2.2.1.2.21. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Female Subjects <sup>4</sup>
- 14.2.2.1.2.22. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) 4
- 14.2.2.1.2.23. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Male Subjects <sup>4</sup>
- 14.2.2.1.2.24. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Female Subjects <sup>4</sup>
- 14.2.2.1.2.25. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) 4
- 14.2.2.1.2.26. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Male Subjects <sup>4</sup>
- 14.2.2.1.2.27. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Female Subjects <sup>4</sup>
- 14.2.2.1.2.28. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) <sup>4</sup>
- 14.2.2.1.2.29. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma

Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Male Subjects <sup>4</sup>

14.2.2.1.2.30. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Concentrations Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Female Subjects <sup>4</sup>

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

<sup>4</sup> To be generated as follows:

| Cubicat No. | | | Pre-Dose | | | | T | ime Post-Da | ay 13 Dose | (h) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject No. | Day 9 | Day 10 | Day 11 | Day 12 | Day 13 | X.XX | Z.ZZ | ZZ.Z | X.XX | X.XX | X.XX |
| <subject id=""></subject> | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| <insert as="" deemed="" many="" n<="" rows="" td=""><td>ecessary&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></insert> | ecessary> | | | | | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Gmean ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GSD ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Gmean 95% CI Upper ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean 95% CI Lower ( <umitsc>)</umitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean 95% CI Upper ( mits ) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum ( <unitsc>)</unitsc> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

n – Number of Subjects; Gmean – Geometric Mean; Amean – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

BLQ - Below the Limit of Quantification (LLOQ = <LLOQ> <unitsC>) of the assay (taken as missing for the calculation of log-transformed statistics and as zero for the calculation of the remaining summary statistics)

ND - Not Done

Program: <SAS Program>



#### 14.2.2.1.3. Plasma Pharmacokinetic Parameters

- 14.2.2.1.3.1. Givinostat: Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1)<sup>3</sup>
- 14.2.2.1.3.2. Givinostat: Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.3.3. Givinostat: Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.1.3.4. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.1.3.5. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.3.6. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.1.3.7. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.1.3.8. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.3.9. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.1.3.10. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) <sup>3</sup>
- 14.2.2.1.3.11. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.1.3.12. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>



14.2.2.1.3.13. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) <sup>3</sup>

14.2.2.1.3.14. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects <sup>3</sup>

14.2.2.1.3.15. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects <sup>4</sup>

4 To be generated as follows:

| Subject No. | C <sub>max</sub><br>( <unitsc>)</unitsc> | T <sub>max</sub> (h) | AUC <sub>0-t</sub><br>( <unitsa>)</unitsa> | AUC <sub>0∞</sub><br>( <unitsa>)</unitsa> | %AUC <sub>extrap</sub><br>(%) | λ <sub>z</sub><br>(1/h) | (h) |
|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| <insert as="" many="" rows<="" td=""><td>as deemed nec</td><td>essary&gt;</td><td></td><td></td><td></td><td></td><td></td></insert> | as deemed nec | essary> | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Gmean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |

n – Number of Subjects; Gmean – Geometric Mean; Amean – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

NC - Not Calculated Program: <SAS Program>



# 14.2.2.1.3.16. Plasma Metabolic Ratios for Givinostat Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) Following Single-Dose Administration of Givinostat (Day 1)

| Subject No. | ITF2374 | ITF2375 | ITF2440 | ITF2563 |
|---|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | XX.XX | XX.XX |
| <insert as="" d<="" many="" rows="" td=""><td>eemed necessary&gt;</td><td></td><td></td><td></td></insert> | eemed necessary> | | | |
| n | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX |
| Gmean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX |

n - Number of Subjects; Gmean - Geometric Mean; Amean - Arithmetic Mean; GSD - Geometric Standard Deviation; SD - Standard Deviation; GCV% - Geometric Coefficient of Variation; CV% - Coefficient of Variation; Gmean 95% CI Lower - Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper - Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower - Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper - Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

NC - Not Calculated

Program: <SAS Program>



- 14.2.2.1.3.17. Givinostat: Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.1.3.18. Givinostat: Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>4</sup>
- 14.2.2.1.3.19. Givinostat: Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>4</sup>
- 14.2.2.1.3.20. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.1.3.21. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>4</sup>
- 14.2.2.1.3.22. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>4</sup>
- 14.2.2.1.3.23. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.1.3.24. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>4</sup>
- 14.2.2.1.3.25. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects <sup>4</sup>
- 14.2.2.1.3.26. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.1.3.27. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>4</sup>
- 14.2.2.1.3.28. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>4</sup>
- 14.2.2.1.3.29. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.1.3.30. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma

Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects <sup>4</sup>

14.2.2.1.3.31. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects <sup>4</sup>

4 To be generated as follows:

| Subject No. | C <sub>max,55</sub><br><unitsc>)</unitsc> | T <sub>max,55</sub> (h) | AUC <sub>0-7,55</sub><br>( <unitsa>)</unitsa> | AUC <sub>0-t</sub><br>( <unitsa>)</unitsa> | AUC <sub>0-∞</sub><br>( <unitsa>)</unitsa> | λ <sub>z</sub><br>(1/h) | t <sub>1/2</sub><br>(h) | CL <sub>ss</sub> /F<br>(L/h) | V <sub>D</sub> /F<br>(L) |
|---|---|---|---|---|---|---|---|---|---|
| <subject<br>ID&gt;</subject<br> | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | x.xxx | XX.XX | XX.XX | XX.XX |
| <insert as="" man<="" td=""><td>ny rows as de</td><td>eemed ne</td><td>cessary&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td></insert> | ny rows as de | eemed ne | cessary> | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| CI Lower | | | | | | | | | |
| Gmean 95% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| CI Upper | | | | | | | | | |
| Amean 95% | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| CI Lower | | | | | | | | | |
| Amean 95% | XX.XX | XX,XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| CI Upper | | | | | | | | | |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX | XX.XX | XX.XX |

n - Number of Subjects; Gmean - Geometric Mean; Amean - Arithmetic Mean; GSD - Geometric Standard Deviation; SD - Standard Deviation; GCV% - Geometric Coefficient of Variation; CV% - Coefficient of Variation; Gmean 95% CI Lower - Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper - Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower - Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper - Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

NC - Not Calculated Program: <SAS Program>

- 14.2.2.1.3.32. Givinostat: Individual Data and Descriptive Statistics of Accumulation Index 4
- 14.2.2.1.3.33. Givinostat: Individual Data and Descriptive Statistics of Accumulation Index Male Subjects <sup>4</sup>
- 14.2.2.1.3.34. Givinostat: Individual Data and Descriptive Statistics of Accumulation Index Female Subjects <sup>4</sup>
- 14.2.2.1.3.35. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Accumulation Index 4
- 14.2.2.1.3.36. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Accumulation Index Male Subjects <sup>4</sup>
- 14.2.2.1.3.37. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Accumulation Index Female Subjects <sup>4</sup>
- 14.2.2.1.3.38. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Accumulation Index <sup>4</sup>
- 14.2.2.1.3.39. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Accumulation Index Male Subjects <sup>4</sup>
- 14.2.2.1.3.40. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Accumulation Index Female Subjects <sup>4</sup>
- 14.2.2.1.3.41. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Accumulation Index 4
- 14.2.2.1.3.42. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Accumulation Index Male Subjects <sup>4</sup>
- 14.2.2.1.3.43. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Accumulation Index Female Subjects <sup>4</sup>
- 14.2.2.1.3.44. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Accumulation Index ⁴
- 14.2.2.1.3.45. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Accumulation Index Male Subjects <sup>4</sup>
- 14.2.2.1.3.46. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Accumulation Index Female Subjects <sup>4</sup>

4 To be generated as follows:

| Subject No. | C <sub>max</sub> | AUC |
|---|---|---|
| <subject id=""></subject> | XX.XX | xx.xx |
| <insert as="" deemed="" many="" no<="" rows="" th=""><th>ecessary&gt;</th><th></th></insert> | ecessary> | |
| n | XX | XX |
| Amean | XX.XX | XX.XX |
| SD | XX.XX | XX.XX |
| SE | XX.X | XX.X |
| Median | XX.XX | XX.XX |
| Minimum | XX XX | XX.XX |
| Maximum | XX.XX | XX.XX |

n - Number of Subjects; Amen - Arithmetic Mean; SD - Standard Deviation; SE - Standard Error.

NC - Not Calculated Program: <SAS Program>



# 14.2.2.1.3.47. Plasma Metabolic Ratios for Givinostat Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) Following Multiple-Dose Administration of Givinostat (Day 13)

| Subject No. | ITF2374 | ITF2375 | ITF2440 | ITF2563 |
|---|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | xx.xx | xx.xx |
| <insert as="" d<="" many="" rows="" td=""><td>eemed necessary&gt;</td><td></td><td></td><td></td></insert> | eemed necessary> | | | |
| n | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX |
| Gmean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX |
| Amean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX |

n – Number of Subjects; Gmeen – Geometric Mean; Ameen – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmeen 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmeen 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Geometric Mean; Ameen 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Ameen 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

NC - Not Calculated Program: <SAS Program>

### 14.2.2.1.4. Log-Linear Regression Parameters for λ<sub>z</sub> Estimation

- 14.2.2.1.4.1. Givinostat: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Single-Dose Administration of Givinostat (Day 1) <sup>6</sup>
- 14.2.2.1.4.2. Givinostat Metabolite (ITF2374): Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Single-Dose Administration of Givinostat (Day 1) <sup>6</sup>
- 14.2.2.1.4.3. Givinostat Metabolite (ITF2375): Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Single-Dose Administration of Givinostat (Day 1) <sup>6</sup>
- 14.2.2.1.4.4. Givinostat Metabolite (ITF2440): Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Single-Dose Administration of Givinostat (Day 1) <sup>6</sup>
- 14.2.2.1.4.5. Givinostat Metabolite (ITF2563): Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Single-Dose Administration of Givinostat (Day 1) <sup>6</sup>
- 14.2.2.1.4.6. Givinostat: Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Multiple-Dose Administration of Givinostat (Day 13) <sup>6</sup>
- 14.2.2.1.4.7. Givinostat Metabolite (ITF2374): Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Multiple-Dose Administration of Givinostat (Day 13) <sup>6</sup>
- 14.2.2.1.4.8. Givinostat Metabolite (ITF2375): Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Multiple-Dose Administration of Givinostat (Day 13) <sup>6</sup>
- 14.2.2.1.4.9. Givinostat Metabolite (ITF2440): Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Multiple-Dose Administration of Givinostat (Day 13) <sup>6</sup>
- 14.2.2.1.4.10. Givinostat Metabolite (ITF2563): Log-Linear Regression Parameters for  $\lambda_z$  Estimation Following Multiple-Dose Administration of Givinostat (Day 13) <sup>6</sup>

6 To be generated as follows:

| Subject No. | Lower TLIN<br>(h) | Upper TLIN (h) | No. of Time Points | RSQ |
|---|---|---|---|---|
| <subject id=""></subject> | xx.xx | xx.xx | xx | x.xx |

#### <Insert as many rows as deemed necessary>

Lower TLIN - Lower Time Point Used in Regression Analysis; Upper TLIN - Upper Time Point Used in Regression Analysis; RSQ - Goodness of Fit for the Terminal Elimination Phase

Program: <SAS Program>

## 14.2.2.2. Urinary Pharmacokinetic Data

## 14.2.2.2.1. Deviations from Urine Sampling Schedule

## 14.2.2.2.1.1. Missing Urine Samples

| Subject No. | Day of<br>Dose | Planned Start Time<br>(h:min) | Planned End Time<br>(h:min) | Reason for Missing Urine Sample |
|---|---|---|---|---|
| <subject id=""></subject> | <day #=""></day> | <planned blood="" sampling="" time=""></planned> | <planned blood="" sampling="" time=""></planned> | <reason blood="" for="" missing="" sample=""></reason> |
| <insert as<br="">many rows as<br/>deemed<br/>necessary&gt;</insert> | | | | |

Program: <SAS Program>



#### 14.2.2.2.2. Urinary Excretion Profile

- 14.2.2.2.1. Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.2.2. Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.3. Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.2.4. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.2.5. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.6. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.2.7. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.2.8. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.9. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.2.2.10. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.2.2.11. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.2.12. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.2.2.13. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.2.2.14. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.15. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>



- 14.2.2.2.16. Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) 3
- 14.2.2.2.17. Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.18. Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.2.2.19. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) <sup>3</sup>
- 14.2.2.2.2.0. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.2.1. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.2.2.2. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) <sup>3</sup>
- 14.2.2.2.2.3. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.2.4. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>
- 14.2.2.2.25. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) $^3$
- 14.2.2.2.2.6. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>3</sup>
- 14.2.2.2.2.7. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>3</sup>

14.2.2.2.28. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) 3

14.2.2.2.2.9. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects <sup>3</sup>

14.2.2.2.30. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects <sup>3</sup>

4 To be generated as follows:

| CALLAN | Pre-Dose | | | Post-Da | y 1 Dose | | |
|---|---|---|---|---|---|---|---|
| Subject No. | (Day -1) | 0h - 12h | 12h - 24h | 24h - 36h | 36h – 48h | 48h - 72h | 72h – 96h |
| <subject id=""></subject> | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| <insert as="" deemed<="" many="" rows="" td=""><td>necessary&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td></insert> | necessary> | | | | | | |
| n | XX | XX | XX | XX | XX | XX | XX |
| Gmean ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean (amits) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| GSD ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| SD ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower ( units ) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Gmean 95% CI Upper ( units ) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean 95% CI Lower ( units ) | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean 95% CI Upper ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Median ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | x.xxx | XX.XX |
| Minimum ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Maximum ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | x.xxx | XX.XX |

n – Number of Subjects; Gmean – Geometric Mean; Amean – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

ND – Not Done

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- 14.2.2.2.31. Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) 3
- 14.2.2.2.32. Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.33. Givinostat: Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>
- 14.2.2.2.34. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) 3
- 14.2.2.2.35. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.36. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>
- 14.2.2.2.37. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) 3
- 14.2.2.2.38. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.39. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>
- 14.2.2.2.2.40. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) 3
- 14.2.2.2.2.41. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.42. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>
- 14.2.2.2.2.43. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) 3
- 14.2.2.2.2.44. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.45. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>



- 14.2.2.2.2.46. Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) <sup>3</sup>
- 14.2.2.2.47. Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.48. Givinostat: Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>
- 14.2.2.2.2.49. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) <sup>3</sup>
- 14.2.2.2.50. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.51. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>
- 14.2.2.2.52. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) <sup>3</sup>
- 14.2.2.2.53. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.54. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>
- 14.2.2.2.55. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) <sup>3</sup>
- 14.2.2.2.56. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>3</sup>
- 14.2.2.2.57. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>3</sup>

14.2.2.2.58. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) 3

14.2.2.2.59. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects <sup>3</sup>

14.2.2.2.2.60. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Cumulative Amount Urinary Excretion Profile Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects <sup>3</sup>

4 To be generated as follows:

| | | | Post-Day | 13 Dose | | |
|---|---|---|---|---|---|---|
| Subject No. | 0h-12h | 12h - 24h | 24h - 36h | 36h - 48h | 48h - 72h | 72h – 96h |
| <subject id=""></subject> | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| <insert as="" deemed="" many="" necessary="" rows=""></insert> | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Gmean ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean (qunits>) | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| GSD ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| SD ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower (units) | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Gmean 95% CI Upper ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean 95% CI Lower ( mits ) | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Amean 95% CI Upper ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |
| Median ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | x.xxx | XX.XX |
| Minimum ( <units>)</units> | XX.XX | XX.XX | XX.XX | XX.XX | x.xxx | XX.XX |
| Maximum (\cunits>) | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX | XX.XX |

n – Number of Subjects; Gmean – Geometric Mean; Amean – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

ND - Not Done

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### 14.2.2.2.3. Urinary Pharmacokinetic Parameters

- 14.2.2.2.3.1. Givinostat: Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) 4
- 14.2.2.3.2. Givinostat: Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>4</sup>
- 14.2.2.2.3.3. Givinostat: Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>4</sup>
- 14.2.2.2.3.4. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) 4
- 14.2.2.2.3.5. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>4</sup>
- 14.2.2.2.3.6. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>4</sup>
- 14.2.2.2.3.7. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) <sup>4</sup>
- 14.2.2.2.3.8. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>4</sup>
- 14.2.2.2.3.9. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>4</sup>
- 14.2.2.2.3.10. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) <sup>4</sup>
- 14.2.2.2.3.11. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Male Subjects <sup>4</sup>
- 14.2.2.2.3.12. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) Female Subjects <sup>4</sup>



14.2.2.2.3.13. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) 4

14.2.2.2.3.14. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Male Subjects <sup>4</sup>

14.2.2.3.15. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) – Female Subjects <sup>4</sup>

4 To be generated as follows:

| Subject No. | R <sub>max</sub><br>( <units>)</units> | tu <sub>max</sub><br>(h) | Amtcum<br>( <units>)</units> | AURC <sub>0-t</sub><br>( <units>)</units> | REC%<br>(%) | CL <sub>R</sub> /F<br>(L/h) |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | x.xxx |
| <insert as="" many="" rows<="" td=""><td>as deemed neces</td><td>sary&gt;</td><td></td><td></td><td></td><td></td></insert> | as deemed neces | sary> | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX.XX | XX.XX | XX,XX | X.XXX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX | XX,XX | X.XXX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Gmean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Amean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Amean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |

n - Number of Subjects; Gmean - Geometric Mean; Amean - Arithmetic Mean; GSD - Geometric Standard Deviation; SD - Standard Deviation; GCV% - Geometric Coefficient of Variation; CV% - Coefficient of Variation; Gmean 95% CI Lower - Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper - Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower - Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper - Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

NC - Not Calculated Program: <SAS Program>

14.2.2.2.3.16. Percentage of Dose Recovered in Urine for Givinostat and Givinostat Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) Following Single-Dose Administration of Givinostat (Day 1)

| Subject No. | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563 | Total |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX |
| <insert as="" many<="" td=""><td>rows as deemed n</td><td>ecessary&gt;</td><td></td><td></td><td></td><td></td></insert> | rows as deemed n | ecessary> | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX XX | XX.XX | XX.XX | XX.XX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| G <sub>mean</sub> 95% CI | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Lower<br>G <sub>mean</sub> 95% CI<br>Upper | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> 95% CI<br>Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> 95% CI<br>Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

n – Number of Subjects; Gmean – Geometric Mean; Amean – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

Total corresponds to the sum of percentage of dose recovered in urine for all analytes

NC - Not Calculated Program: <SAS Program>



- 14.2.2.2.3.17. Givinostat: Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.2.3.18. Givinostat: Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>4</sup>
- 14.2.2.2.3.19. Givinostat: Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>4</sup>
- 14.2.2.2.3.20. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.2.3.21. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>4</sup>
- 14.2.2.3.22. Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>4</sup>
- 14.2.2.2.3.23. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.2.3.24. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>4</sup>
- 14.2.2.2.3.25. Givinostat Metabolite (ITF2375): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>4</sup>
- 14.2.2.2.3.26. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) 4
- 14.2.2.3.27. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Male Subjects <sup>4</sup>
- 14.2.2.2.3.28. Givinostat Metabolite (ITF2440): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) Female Subjects <sup>4</sup>

14.2.2.2.3.29. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) <sup>4</sup>

14.2.2.2.3.30. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Male Subjects <sup>4</sup>

14.2.2.3.31. Givinostat Metabolite (ITF2563): Individual Data and Descriptive Statistics of Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) – Female Subjects <sup>4</sup>

4 To be generated as follows:

| Subject No. | R <sub>max</sub><br>( <units>)</units> | tu <sub>max</sub><br>(h) | Amtcum<br>( <units>)</units> | AURC <sub>0-t</sub><br>( <units>)</units> | REC%<br>(%) | CL <sub>R</sub> /F<br>(L/h) |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | xx.xx | XX.XX | xx.xx | xx.xx | xx.xx | x.xxx |
| <insert as="" many="" rows<="" td=""><td>as deemed neces</td><td>sary&gt;</td><td></td><td></td><td></td><td></td></insert> | as deemed neces | sary> | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Gmean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Gmean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Amean 95% CI Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Amean 95% CI Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | X.XXX |

n - Number of Subjects; Gmean - Geometric Mean; Amean - Arithmetic Mean; GSD - Geometric Standard Deviation; SD - Standard Deviation; GCV% - Geometric Coefficient of Variation; CV% - Coefficient of Variation; Gmean 95% CI Lower - Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper - Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower - Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper - Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

NC - Not Calculated

Program: <SAS Program>

14.2.2.2.3.32. Percentage of Dose Recovered in Urine for Givinostat and Givinostat Metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) Following Multiple-Dose Administration of Givinostat (Day 13)

| Subject No. | Givinostat | ITF2374 | ITF2375 | ITF2440 | ITF2563 | Total |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| <insert as="" many<="" td=""><td>rows as deemed n</td><td>ecessary&gt;</td><td></td><td></td><td></td><td></td></insert> | rows as deemed n | ecessary> | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Gmean | XX.XX | XX.XX | XX XX | XX.XX | XX.XX | XX.XX |
| Amean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GSD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| GCV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| G <sub>mean</sub> 95% CI<br>Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| G <sub>mean</sub> 95% CI<br>Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> 95% CI<br>Lower | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| A <sub>mean</sub> 95% CI<br>Upper | XX.XX | XX.XX | XX.XX | XX.XX | XX XX | XX.XX |
| Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

n – Number of Subjects; Gmean – Geometric Mean; Amean – Arithmetic Mean; GSD – Geometric Standard Deviation; SD – Standard Deviation; GCV% – Geometric Coefficient of Variation; CV% – Coefficient of Variation; Gmean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Geometric Mean; Gmean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Geometric Mean; Amean 95% CI Lower – Lower Limit of the 95% Confidence Interval for the Arithmetic Mean; Amean 95% CI Upper – Upper Limit of the 95% Confidence Interval for the Arithmetic Mean.

Total corresponds to the sum of percentage of dose recovered in urine for all analytes

NC - Not Calculated Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- 14.2.2.3. Plasma Concentration Versus Time Profiles of All Subjects
- 14.2.2.3.1. Givinostat: Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) – Linear Scale
- 14.2.2.3.2. Givinostat: Plasma Concentration *Versus* Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) – Linear Scale
- 14.2.2.3.3. Givinostat Metabolite (ITF2374): Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) Linear Scale
- 14.2.2.3.4. Givinostat Metabolite (ITF2374): Plasma Concentration Versus Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) Linear Scale
- 14.2.2.3.5. Givinostat Metabolite (ITF2375): Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) Linear Scale
- 14.2.2.3.6. Givinostat Metabolite (ITF2375): Plasma Concentration Versus Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) Linear Scale
- 14.2.2.3.7. Givinostat Metabolite (ITF2440): Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) Linear Scale
- 14.2.2.3.8. Givinostat Metabolite (ITF2440): Plasma Concentration *Versus* Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) Linear Scale
- 14.2.2.3.9. Givinostat Metabolite (ITF2563): Plasma Concentration Versus Time Profiles of All Subjects Following Single-Dose Administration of Givinostat (Day 1) Linear Scale
- 14.2.2.3.10. Givinostat Metabolite (ITF2563): Plasma Concentration Versus Time Profiles of All Subjects Following Multiple-Dose Administration of Givinostat (Day 13) Linear Scale



Clinical Study Report

#### 14.2.2.4. Individual Plasma Concentration Versus Time Profiles

- 14.2.2.4.1. Givinostat: Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale
- 14.2.2.4.2. Givinostat: Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale
- 14.2.2.4.3. Givinostat: Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) - Linear Scale
- 14.2.2.4.4. Givinostat: Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) - Semi-Logarithmic Scale
- 14.2.2.4.5. Givinostat: Individual Trough Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) — Linear Scale
- 14.2.2.4.6. Givinostat Metabolite (ITF2374): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale
- 14.2.2.4.7. Givinostat Metabolite (ITF2374): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Semi-Logarithmic Scale
- 14.2.2.4.8. Givinostat Metabolite (ITF2374): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale
- 14.2.2.4.9. Givinostat Metabolite (ITF2374): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) — Semi-Logarithmic Scale
- 14.2.2.4.10. Givinostat Metabolite (ITF2374): Individual Trough Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) - Linear Scale
- 14.2.2.4.11. Givinostat Metabolite (ITF2375): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale
- 14.2.2.4.12. Givinostat Metabolite (ITF2375): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat — Semi-Logarithmic Scale
- 14.2.2.4.13. Givinostat Metabolite (ITF2375): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale
- 14.2.2.4.14. Givinostat Metabolite (ITF2375): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) — Semi-Logarithmic Scale
- 14.2.2.4.15. Givinostat Metabolite (ITF2375): Individual Trough Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) – Linear Scale



- 14.2.2.4.16. Givinostat Metabolite (ITF2440): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.4.17. Givinostat Metabolite (ITF2440): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Semi-Logarithmic Scale
- 14.2.2.4.18. Givinostat Metabolite (ITF2440): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale
- 14.2.2.4.19. Givinostat Metabolite (ITF2440): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Semi-Logarithmic Scale
- 14.2.2.4.20. Givinostat Metabolite (ITF2440): Individual Trough Plasma Concentration *Versus* Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale
- 14.2.2.4.21. Givinostat Metabolite (ITF2563): Individual Plasma Concentration Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.4.22. Givinostat Metabolite (ITF2563): Individual Plasma Concentration *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Semi-Logarithmic Scale
- 14.2.2.4.23. Givinostat Metabolite (ITF2563): Individual Plasma Concentration Versus Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale
- 14.2.2.4.24. Givinostat Metabolite (ITF2563): Individual Plasma Concentration *Versus* Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Semi-Logarithmic Scale
- 14.2.2.4.25. Givinostat Metabolite (ITF2563): Individual Trough Plasma Concentration *Versus* Time Profile Following Multiple-Dose Administration of Givinostat (Day 9 to Day 13) Linear Scale



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

- 14.2.2.5. Individual Urinary Excretion Versus Time Profiles
- 14.2.2.5.1. Givinostat: Individual Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.2. Givinostat: Individual Cumulative Amount Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.3. Givinostat Metabolite (ITF2374): Individual Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.4. Givinostat Metabolite (ITF2374): Individual Cumulative Amount Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.5. Givinostat Metabolite (ITF2375): Individual Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.6. Givinostat Metabolite (ITF2375): Individual Cumulative Amount Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.7. Givinostat Metabolite (ITF2440): Individual Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.8. Givinostat Metabolite (ITF2440): Individual Cumulative Amount Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.9. Givinostat Metabolite (ITF2563): Individual Urinary Excretion *Versus* Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat Linear Scale
- 14.2.2.5.10. Givinostat Metabolite (ITF2563): Individual Cumulative Amount Urinary Excretion Versus Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale

Version: <Version>
Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### 14.2.3. SAFETY DATA - PART 3

#### 14.2.3.1. Adverse Events

#### 14.2.3.1.1. Pre-Treatment Adverse Events

| Subject No. | SOC | SAE? Adverse Ev | | t Date and Time | Maximal | C P | Medication | |
|---|---|---|---|---|---|---|---|---|
| | MedDRA PT<br>(Reported Term) | (Yes/No) | Start | End | Severity | Causality | Required? | Outcome |
| <subject id=""></subject> | <soc> <teae in="" meddra="" pt=""> (<teae reported="" term="">)</teae></teae></soc> | <yes no=""></yes> | DDMMMYYYY<br>hh:mm> | -DDMMMYYYY-<br>hh mm> | <maximal<br>Severity of the<br/>AE&gt;</maximal<br> | <causality of<br="">the AE&gt;</causality> | <yes no=""></yes> | <outcome of<br="">the AE&gt;</outcome> |

<Insert as many rows as deemed necessary>

SOC - System Organ Class; MedDRA - Medical Dictionary for Regulatory Activities; PT - Preferred Term; SAE - Serious Adverse Event NK - Not Known

Program: <SAS Program>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

#### 14.2.3.1.2. Treatment-Emergent Adverse Events (I)

| Cubicat No. | Day of Doss | SOC<br>MedDRA PT | SAE? | Last Treatment | Adverse Event Date and Time | |
|---|---|---|---|---|---|---|
| Subject No. | Day of Dose | (Reported Term) | (Yes/No) | Date and Time | Start | Start |
| <subject id=""></subject> | <day#></day#> | <soc> <teae in="" meddra="" pt=""> (<teae reported="" term="">)</teae></teae></soc> | <yes no=""></yes> | <ddmmmyyyy hh="" mm=""></ddmmmyyyy> | <ddmmmyyyy hh:mm=""></ddmmmyyyy> | <ddmmmyyyy hh:mm=""></ddmmmyyyy> |

<Insert as many rows as deemed necessary>

SOC - System Organ Class; MedDRA - Medical Dictionary for Regulatory Activities; PT - Preferred Term; SAE - Serious Adverse Event

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

## 14.2.3.1.3. Treatment-Emergent Adverse Events (II)

| Subject No. | Day of Dose | SOC<br>MedDRA PT<br>(Reported Term) | Maximal Severity | Causality | Medication<br>Required? | Outcome |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | <day #=""></day> | <soc> <teae in="" meddra="" pt=""> (<teae reported="" term="">)</teae></teae></soc> | <maximal of="" severity="" teae="" the=""></maximal> | <causality of="" the<br="">TEAE&gt;</causality> | <yes no=""></yes> | <outcome of="" teae="" the=""></outcome> |

<Insert as many rows as deemed necessary>

SOC - System Organ Class; MedDRA - Medical Dictionary for Regulatory Activities; PT - Preferred Term; SAE - Serious Adverse Event

Program: <SAS Program>

- 14.2.3.2. Vital Signs
- 14.2.3.2.1. Descriptive Statistics of Vital Signs Parameters 9
- 14.2.3.2.2. Descriptive Statistics of Change from Baseline of Vital Signs Parameters 9
- 14.2.3.2.3. Shifts in Vital Signs Parameters 10
- 14.2.3.3. 12-Lead ECG
- 14.2.3.3.1. Descriptive Statistics of 12-Lead ECG Parameters 9
- 14.2.3.3.2. Descriptive Statistics of Change from Baseline of 12-Lead ECG Parameters 9
- 14.2.3.3.3. Shifts in 12-Lead ECG Parameters 10
- 14.2.3.4. Hematology
- 14.2.3.4.1. Descriptive Statistics of Hematology Parameters 9
- 14.2.3.4.2. Descriptive Statistics of Change from Baseline of Hematology Parameters 9
- 14.2.3.4.3. Shifts in Hematology Parameters 10
- 14.2.3.5. Biochemistry
- 14.2.3.5.1. Descriptive Statistics of Biochemistry Parameters 9
- 14.2.3.5.2. Descriptive Statistics of Change from Baseline of Biochemistry Parameters 9
- 14.2.3.5.3. Shifts in Biochemistry Parameters 10
- 14.2.3.6. Coagulation
- 14.2.3.6.1. Descriptive Statistics of Coagulation Parameters 9
- 14.2.3.6.2. Descriptive Statistics of Change from Baseline of Coagulation Parameters 9
- 14.2.3.6.3. Shifts in Coagulation Parameters 10
- 14.2.3.7. Urinalysis
- 14.2.3.7.1. Descriptive Statistics of Urinalysis Parameters 9
- 14.2.3.7.2. Descriptive Statistics of Change from Baseline of Urinalysis Parameters 9

## 14.2.3.7.3. Shifts in Urinalysis Parameters 10

## 9 To be generated as follows:

| Parameter | Study Day | Protocol Time | n | Mean | SD | SE | Median | Minimum | Maximum |
|---|---|---|---|---|---|---|---|---|---|
| <parameter (unit)=""><day></day></parameter> | | <protocol time=""> <protocol time=""> <protocol time=""> <protocol time=""></protocol></protocol></protocol></protocol> | XX | X.XXX | X.XXX | X.XXX | x.xxx | x.xxx | x.xxx |
| <insert as="" man<="" td=""><td>y rows as deemed ne</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></insert> | y rows as deemed ne | | | | | | | | |

n - number of subjects; SD - Standard Deviation; SE - Standard Error

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

10 To be generated as follows:

| | 5 × 1 × 2 × | | Class | | |
|---|---|---|---|---|---|
| Parameter | Study Day | Protocol Time | Baseline | Post-Baseline<br>Assessment | Nr. of Subjects |
| <parameter (un<="" td=""><td>it)&gt; <day></day></td><td><protocol time=""></protocol></td><td><low <br="">Normal/<br/>High&gt;</low></td><td><low <br="">Normal/<br/>High&gt;</low></td><td>xx</td></parameter> | it)> <day></day> | <protocol time=""></protocol> | <low <br="">Normal/<br/>High&gt;</low> | <low <br="">Normal/<br/>High&gt;</low> | xx |
| | | <protocol time=""></protocol> | <low <br="">Normal/<br/>High&gt;</low> | <low <br="">Normal/<br/>High&gt;</low> | XX |
| <insert as="" many<="" td=""><td>rows as deemed ne</td><td>cessary&gt;</td><td></td><td></td><td></td></insert> | rows as deemed ne | cessary> | | | |

Program: SAS Program
14.2.3.8. Body Weight

14.2.3.8.1. Descriptive Statistics of Body Weight 9

14.2.3.8.2. Descriptive Statistics of Body Weight - Male Subjects 9

14.2.3.8.3. Descriptive Statistics of Body Weight - Female Subjects 9

14.2.3.8.4. Descriptive Statistics of Change from Baseline of Body Weight 9

14.2.3.8.5. Descriptive Statistics of Change from Baseline of Body Weight - Male Subjects 9

14.2.3.8.6. Descriptive Statistics of Change from Baseline of Body Weight - Female Subjects 9

# 9 To be generated as follows:

| | Mean | SD | SE | Median | Minimum | Maximum |
|---|---|---|---|---|---|---|
| xx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx | x.xxx |
| | XX | xx x.xxx<br>deemed necessary> | | The state of the s | THE STREET STREET | |

n - number of subjects; SD - Standard Deviation; SE - Standard Error

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

A.4. List of Subject Data Listings (Section 16.2 of CSR)

A.4.1. Part 3

16.2.1. PART 3

16.2.1.1. Subject Disposition

16.2.1.1.1. Subject Disposition

| Screening<br>No. | Date ICF Signed | Subject<br>Eligible? | Subject Given<br>an Unique<br>Subject No.? | Unique Subject No. | Inclusion Criteria<br>Not Met | Exclusion Criteria<br>Met | Other Reason for<br>Non-Eligibility | Reason for<br>Non-<br>Randomization |
|---|---|---|---|---|---|---|---|---|
| <screening<br>number&gt;</screening<br> | <ddmmmyyyy< td=""><td>&gt;<yes no=""></yes></td><td><yes no=""></yes></td><td><unique subject<br="">No&gt;</unique></td><td><list all="" inclusion<br="">criteria that were<br/>not met&gt;</list></td><td></td><td></td><td><ul> <li>List reason for<br/>non-randomization</li> </ul></td></ddmmmyyyy<> | > <yes no=""></yes> | <yes no=""></yes> | <unique subject<br="">No&gt;</unique> | <list all="" inclusion<br="">criteria that were<br/>not met&gt;</list> | | | <ul> <li>List reason for<br/>non-randomization</li> </ul> |
| <insert as="" m<="" td=""><td>any rows as deemed</td><td>necessary&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td></insert> | any rows as deemed | necessary> | | | | | | |

ICF - Informed Consent Form Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.2. Protocol Deviations

# 16.2.1.2.1. Blood Sampling Times Deviations

| Cubicat No. | Campling Timenaint | Sampling Da | ate and Time | —Deviation Reason |
|---|---|---|---|---|
| Subject No. | Sampling Timepoint | Scheduled/Target | Actual | —Deviation Keason |
| <subject id=""></subject> | <scheduled or="" time="" unscheduled=""></scheduled> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <reason deviation="" for=""></reason> |
| <insert as="" many="" rows<="" td=""><td>s as deemed necessary&gt;</td><td></td><td></td><td></td></insert> | s as deemed necessary> | | | |

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

### 16.2.1.2.2. Other Protocol Deviations

| Subject No. Protocol<br>Phase | Category | Description | Classification |
|---|---|---|---|
| Subject ID> <protocol<br>Phase #&gt;</protocol<br> | <deviation<br>Category&gt;</deviation<br> | <description deviation="" of="" the=""></description> | <pre><important important="" not=""></important></pre> |

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.3. Excluded Data from the Pharmacokinetic Analysis

#### 16.2.1.3.1. Plasma Concentrations

#### 16.2.1.3.1.1. Individual Data of Plasma Concentrations

| Subject No. Day of Dosing Analyte | | | Des David | | | | | Time Po | st-Dose (h) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject No | Dosing | Analyte | Pre-dose | X.XX | Z.ZZ | X.XX | ZZ.ZZ | X.XX | Z.ZZ | X.XX | 7.77 | X.XX | 7.77 |
| <subject< td=""><td><day #=""></day></td><td><analyte></analyte></td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td><td>XX.XX</td></subject<> | <day #=""></day> | <analyte></analyte> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

<Insert as many rows as deemed necessary>

BLQ - Below the Limit of Quantification (LLOQ = <LLOQ> <unitsC>) of the assay

ND - Not Done

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

### 16.2.1.3.2. Plasma Concentration Versus Time Profiles

#### 16.2.1.3.2.1. Individual Plasma Concentration Versus Time Profiles - Linear Scale

# 16.2.1.3.2.2. Individual Plasma Concentration Versus Time Profiles - Semi-Logarithmic Scale

Note: These Figures will be extracted from Phoenix® WinNonlin® 8.2 or higher. A figure will be produced for each subject with data excluded from the pharmacokinetic analysis.



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.3.3. Urine Excretion

#### 16.2.1.3.3.1. Individual Data of Plasma Concentrations

| | Day of | 6 6 3 | | | | Time Pos | t-Dose (h) | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject No | Day of<br>Dosing | Analyte | Pre-dose - | 0h - 12h | 12h – 24h | 24h - 36h | 36h – 48h | 48h - 72h | 72h – 96h |
| <subject id=""></subject> | <day #=""></day> | <analyte></analyte> | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |

<Insert as many rows as deemed necessary>

BLQ - Below the Limit of Quantification (LLOQ = <LLOQ> <unitsC>) of the assay

ND - Not Done

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

### 16.2.1.3.4. Urine Excretion Versus Time Profiles

### 16.2.1.3.4.1. Urine Excretion Versus Time Profiles - Linear Scale

Note: These Figures will be extracted from Phoenix® WinNonlin® 8.2 or higher. A figure will be produced for each subject with data excluded from the pharmacokinetic analysis.



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.4. Demographic and Other Baseline Data

# 16.2.1.4.1. Demographic Data

| (years) | (cm) | (kg) | (kg/m <sup>2</sup> ) |
|---------|------|--------|----------------------|
| XX | xxx | XX.X | XX.X |
| | XX | xx xxx | |

<Insert as many rows as deemed necessary>

ICF - Informed Consent Form; BMI - Body Mass Index; M - Male; F - Female

Program: <SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.4.2. Fertility/Contraception

# 16.2.1.4.2.1. Female Fertility/Contraception

| Subject No. | Childbearing Potential? | If Yes, Birth Control Method | Breast Feeding? | Comments |
|---|---|---|---|---|
| <subject id=""></subject> | <yes no=""></yes> | <birth control="" method=""></birth> | <yes no=""></yes> | <comments></comments> |
| <insert a<="" as="" many="" rows="" td=""><td>s deemed necessary&gt;</td><td></td><td></td><td></td></insert> | s deemed necessary> | | | |

# 16.2.1.4.2.2. Male Fertility/Contraception

| Subject No. | Sexually Active? | Agrees to Use Condom? | Female partner agrees to use a highly effective method of contraception? | Agree not to donate sperm<br>from first dose administration<br>until at least 90 days after the<br>last study drug administration | Comments |
|---|---|---|---|---|---|
| <subject id=""></subject> | <yes no=""></yes> | <yes no=""></yes> | <yes no=""></yes> | <yes no=""></yes> | <comments></comments> |
| <insert as="" many<="" td=""><td>rows as deemed necessa</td><td>ary&gt;</td><td></td><td></td><td></td></insert> | rows as deemed necessa | ary> | | | |

Program: <SAS Program>

ITF/2357/55 Version: <Version> Date: <DDMMMYYYY> PPD

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.4.3. Drugs of Abuse, Ethanol and Cotinine

| Subject No. | Date and Time | Amphetamin | iesBenzodiazepi | nesCocaine | Cannabinoid | ls Opiates | Ethanol | Cotinine |
|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <positive <br="">Negative&gt;</positive> | <positive <br="">Negative&gt;</positive> | <positive <br="">Negative&gt;</positive> | <positive <br="">Negative&gt;</positive> | <positive negative=""></positive> | <positive <br="">Negative&gt;</positive> | <positive negative<="" th=""></positive> |

Program: <SAS Program>

Version: <Version> Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.4.4. Viral Serology at Screening

| Subject No. | Actual Date and Time | Protocol Phase | HIV-1 & HIV-2 | Hepatitis B | Hepatitis C |
|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <protocol phase=""></protocol> | <qualitative value=""></qualitative> | <qualitative value=""></qualitative> | <qualitative td="" value<=""></qualitative> |

HIV - Human Immunodeficiency Virus

Program: <SAS Program>
Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.4.5. Previous and Concomitant Medication

| Cubiant Na | t No. Drug Name [ATC Code] Indication Pharmaceutical Dose (units) Frequency Route | | Dants | Dat | Date and Time |
|---|---|---|---|---|---|
| Subject No. | [ATC Code] Indication | Form Dose (units) Frequency | Koute | Start | End |
| | <generic <therapeuti="" [xxxxxxxx]="" name="">indication&gt;</generic> | <pharmaceutical<dose (units)=""><frequency>Form&gt;</frequency></pharmaceutical<dose> | <route></route> | <ddmmmyyyy></ddmmmyyyy> | <ddmmmyyyy or<br="">Ongoing&gt;</ddmmmyyyy> |

ATC - Anatomical Therapeutic Chemical

NK - Not Known

Program: <SAS Program>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.4.6. SARS-COV-2 Test

| Subject No. | Actual Date | Protocol Phase | Result | If Unscheduled, Reason |
|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy></ddmmmyyyy> | <protocol phase=""></protocol> | <not detectable,="" inconclusive=""></not> | <reason></reason> |

<Insert as many rows as deemed necessary>

Program: SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.5. Compliance

# 16.2.1.5.1. Investigational Product Administration

| Subject No. | Date | Actual<br>Clock Time | Dose (units) | Investigational<br>Product<br>Formulation | Route of<br>Administration | Hands and<br>Mouth Check? | 150 mL of<br>water taken? | Comments |
|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy<br>YY/ N/A&gt;</ddmmmyy<br> | <hh a="" mm="" n=""></hh> | <dose (units)=""></dose> | <formulation></formulation> | <route></route> | <yes a<="" n="" no="" td=""><td>&gt;<yes a<="" n="" no="" td=""><td>&gt; <comments></comments></td></yes></td></yes> | > <yes a<="" n="" no="" td=""><td>&gt; <comments></comments></td></yes> | > <comments></comments> |

N/A - Not Applicable

Program: SAS Program>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 16.2.1.6. Individual Pharmacokinetic Data

### 16.2.1.6.1. Givinostat: Individual Pharmacokinetic Data

### 16.2.1.6.1.1. Givinostat: Individual Drug Plasma Concentration Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.2.1. for single-dose data and 14.3.2.1.2.16. for multiple-dose data'

#### 16.2.1.6.1.2. Givinostat: Individual Plasma Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.3.1. for single-dose data and 14.3.2.1.3.16. for multiple-dose data'

#### 16.2.1.6.1.3. Givinostat: Individual Plasma Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.4.1. to 14.3.2.4.2.'

#### 16.2.1.6.1.4. Givinostat: Individual Urine Excretion Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.2.1. for single-dose data and 14.3.2.2.2.16. for multiple-dose data'

#### 16.2.1.6.1.5. Givinostat: Individual Urine Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.3.1. for single-dose data and 14.3.2.2.3.16. for multiple-dose data'

#### 16.2.1.6.1.6. Givinostat: Individual Urine Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.5.1. to 14.3.2.5.2.'

## 16.2.1.6.1.7. Givinostat: Documentation of Statistical Analysis

16.2.1.6.1.7.1. Givinostat: Plasma Non-Compartmental Analysis Output

16.2.1.6.1.7.2. Givinostat: Plasma Non-Compartmental Analysis Plots

#### 16.2.1.6.1.7.3. Givinostat: Urine Non-Compartmental Analysis Output

Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

### 16.2.1.6.2. Givinostat Metabolite (ITF2374): Individual Pharmacokinetic Data

### 16.2.1.6.2.1. Givinostat Metabolite (ITF2374): Individual Drug Plasma Concentration Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.2.4. for single-dose data and 14.3.2.1.2.19. for multiple-dose data'

### 16.2.1.6.2.2. Givinostat Metabolite (ITF2374): Individual Plasma Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.3.4. for single-dose data and 14.3.2.1.3.19. for multiple-dose data'

### 16.2.1.6.2.3. Givinostat Metabolite (ITF2374): Individual Plasma Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.4.3. to 14.3.2.4.4.'

# 16.2.1.6.2.4. Givinostat Metabolite (ITF2374): Individual Urine Excretion Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.2.4. for single-dose data and 14.3.2.2.2.19. for multiple-dose data'

#### 16.2.1.6.2.5. Givinostat Metabolite (ITF2374): Individual Urine Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.3.4. for single-dose data and 14.3.2.2.3.19, for multiple-dose data'

#### 16.2.1.6.2.6. Givinostat Metabolite (ITF2374): Individual Urine Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.5.3. to 14.3.2.5.4.'

#### 16.2.1.6.2.7. Givinostat Metabolite (ITF2374): Documentation of Statistical Analysis

- 16.2.1.6.2.7.1. Givinostat Metabolite (ITF2374): Plasma Non-Compartmental Analysis Output
- 16.2.1.6.2.7.2. Givinostat Metabolite (ITF2374): Plasma Non-Compartmental Analysis Plots

### 16.2.1.6.2.7.3. Givinostat Metabolite (ITF2374): Urine Non-Compartmental Analysis Output

### 16.2.1.6.3. Givinostat Metabolite (ITF2375): Individual Pharmacokinetic Data

### 16.2.1.6.3.1. Givinostat Metabolite (ITF2375): Individual Drug Plasma Concentration Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.2.7. for single-dose data and 14.3.2.1.2.22. for multiple-dose data'

### 16.2.1.6.3.2. Givinostat Metabolite (ITF2375): Individual Plasma Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.3.7. for single-dose data and 14.3.2.1.3.22. for multiple-dose data'

### 16.2.1.6.3.3. Givinostat Metabolite (ITF2375): Individual Plasma Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.4.5. to 14.3.2.4.6.'

# 16.2.1.6.3.4. Givinostat Metabolite (ITF2375): Individual Urine Excretion Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.2.7. for single-dose data and 14.3.2.2.2.2.2 for multiple-dose data'

#### 16.2.1.6.3.5. Givinostat Metabolite (ITF2375): Individual Urine Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.3.7. for single-dose data and 14.3.2.2.3.22, for multiple-dose data'

#### 16.2.1.6.3.6. Givinostat Metabolite (ITF2375): Individual Urine Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.5.5. to 14.3.2.5.6.'

#### 16.2.1.6.3.7. Givinostat Metabolite (ITF2375): Documentation of Statistical Analysis

16.2.1.6.3.7.1. Givinostat Metabolite (ITF2375): Plasma Non-Compartmental Analysis Output

16.2.1.6.3.7.2. Givinostat Metabolite (ITF2375): Plasma Non-Compartmental Analysis Plots

16.2.1.6.3.7.3. Givinostat Metabolite (ITF2375): Urine Non-Compartmental Analysis Output

### 16.2.1.6.4. Givinostat Metabolite (ITF2440): Individual Pharmacokinetic Data

### 16.2.1.6.4.1. Givinostat Metabolite (ITF2440): Individual Drug Plasma Concentration Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.2.14. for single-dose data and 14.3.2.1.2.28. for multiple-dose data'

### 16.2.1.6.4.2. Givinostat Metabolite (ITF2440): Individual Plasma Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.3.14. for single-dose data and 14.3.2.1.3.28. for multiple-dose data'

### 16.2.1.6.4.3. Givinostat Metabolite (ITF2440): Individual Plasma Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.4.9. to 14.3.2.4.10.'

# 16.2.1.6.4.4. Givinostat Metabolite (ITF2440): Individual Urine Excretion Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.2.14. for single-dose data and 14.3.2.2.2.28. for multiple-dose data'

#### 16.2.1.6.4.5. Givinostat Metabolite (ITF2440): Individual Urine Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.3.14. for single-dose data and 14.3.2.2.3.28. for multiple-dose data'

#### 16.2.1.6.4.6. Givinostat Metabolite (ITF2440): Individual Urine Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.5.9. to 14.3.2.5.10.'

#### 16.2.1.6.4.7. Givinostat Metabolite (ITF2440): Documentation of Statistical Analysis

16.2.1.6.4.7.1. Givinostat Metabolite (ITF2440): Plasma Non-Compartmental Analysis Output

16.2.1.6.4.7.2. Givinostat Metabolite (ITF2440): Plasma Non-Compartmental Analysis Plots

#### 16.2.1.6.4.7.3. Givinostat Metabolite (ITF2440): Urine Non-Compartmental Analysis Output

# 16.2.1.6.5. Givinostat Metabolite (ITF2563): Individual Pharmacokinetic Data

### 16.2.1.6.5.1. Givinostat Metabolite (ITF2563): Individual Drug Plasma Concentration Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.2.7. for single-dose data and 14.3.2.1.2.28. for multiple-dose data'

### 16.2.1.6.5.2. Givinostat Metabolite (ITF2563): Individual Plasma Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.1.3.7. for single-dose data and 14.3.2.1.3.28. for multiple-dose data'

### 16.2.1.6.5.3. Givinostat Metabolite (ITF2563): Individual Plasma Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.4.9. to 14.3.2.4.10.'

# 16.2.1.6.5.4. Givinostat Metabolite (ITF2563): Individual Urine Excretion Data

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.2.7. for single-dose data and 14.3.2.2.2.28. for multiple-dose data'

#### 16.2.1.6.5.5. Givinostat Metabolite (ITF2563): Individual Urine Pharmacokinetic Parameters

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.2.3.5. for single-dose data and 14.3.2.2.3.28. for multiple-dose data'

#### 16.2.1.6.5.6. Givinostat Metabolite (ITF2563): Individual Urine Pharmacokinetic Profiles

Note: The following sentence should be inserted in this section: 'No further information is provided; refer to sections 14.3.2.5.9. to 14.3.2.5.10.'

#### 16.2.1.6.5.7. Givinostat Metabolite (ITF2563): Documentation of Statistical Analysis

16.2.1.6.5.7.1. Givinostat Metabolite (ITF2563): Plasma Non-Compartmental Analysis Output

16.2.1.6.5.7.2. Givinostat Metabolite (ITF2563): Plasma Non-Compartmental Analysis Plots

16.2.1.6.5.7.3. Givinostat Metabolite (ITF2563): Urine Non-Compartmental Analysis Output



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.7. Adverse Event Listings (Each Subject)

# 16.2.1.7.1. Pre-Treatment Adverse Events 7

# 16.2.1.7.2. Treatment-Emergent Adverse Events 7

<sup>7</sup> To be generated as follows:

| Subject No | Day of<br>Dose | Treatment | Reported<br>Term | Serious? | Maximal<br>Severity | Causality | Action<br>Taken | Medication<br>Required? | Outcome | Adverse<br>Event Star<br>Date and<br>Time | Adverse<br>t Event End<br>Date and<br>Time | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <day #=""></day> | <investigational product=""></investigational> | <ae<br>Reported<br/>Term&gt;</ae<br> | <yes no=""></yes> | | <not<br>r Reasonably<br/>Possible or<br/>Reasonably<br/>Possible&gt;</not<br> | | | <fatal, not<br="">Recovered<br/>Not<br/>Resolved,<br/>Recovered<br/>Resolved<br/>with<br/>Sequelae,<br/>Recovering<br/>/ Resolving<br/>or<br/>Unknown&gt;</fatal,> | hh mm> | | <comment< td=""></comment<> |

<Insert as many rows as deemed necessary>

NK - Not Known

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Note: The "Investigational Product" column will only be generated for Table 16.2.3.7.2. If an Adverse Event is related to Medical History, that information will be reported in 'Comments'. The "Comments" column will only be generated if there are reported comments for the adverse events.

Version: <Version> Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.7.3. Serious Adverse Events (I)

| Subject No. | Reported Term | Reason for Seriousness | Details |
|---|---|---|---|
| <subject id=""></subject> | <ae reported="" term=""></ae> | <reason></reason> | <sae details=""></sae> |
| <insert a<="" as="" many="" rows="" td=""><td>is deemed necessary&gt;</td><td></td><td></td><td></td></insert> | is deemed necessary> | | |

Program: <SAS Program>
Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.8. Listings of Laboratory Measurements by Subject

# 16.2.1.8.1. Normal Range of Laboratory Values

| Category | | | | Fe | male | N | <b>Lale</b> | |
|---|---|---|---|---|---|---|---|---|
| | Analyte | Age | Units | LLN | ULN | LLN | ULN | Qualitative |
| <category></category> | <laboratory analyte=""></laboratory> | <age interval=""></age> | <units></units> | | | | | <qualitative<br>Values&gt;</qualitative<br> |

<Insert as many rows as deemed necessary>

LLN - Lower Limit Normal; ULN - Upper Limit Normal

Program: <SAS Program>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.2. Hematology (I)

| Subject No. | Actual Date<br>and Time | Protocol<br>Phase | Hemoglobin<br>(g/dL) | RBC<br>(10^12/L) | Hematocrit<br>(%) | MCV<br>(fL) | MCH<br>(pg) | MCHC<br>(g/dL) | RDW-CV<br>(%) | Total WBC<br>(10^9/L) | If<br>Unschedule<br>d, Reason |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <subject id:<="" td=""><td>&gt;<ddmmmy<br>YYY<br/>lth mm&gt;</ddmmmy<br></td><td><protocol<br>Phase&gt;</protocol<br></td><td>XX</td><td>xx</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>xx</td><td>xx</td><td><reason></reason></td></subject> | > <ddmmmy<br>YYY<br/>lth mm&gt;</ddmmmy<br> | <protocol<br>Phase&gt;</protocol<br> | XX | xx | XX | XX | XX | XX | xx | xx | <reason></reason> |

### <Insert as many rows as deemed necessary>

RBC - Red Blood Cell; MCV - Mean Corpuscular Volume; MCH - Mean Corpuscular Hemoglobin; MCHC - Mean Corpuscular Hemoglobin Concentration; RDW-CV - Coefficient Variation of the Red Cell Distribution Width; WBC - White Blood Cell

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.8.3. Hematology (II)

| | Actual Data | Duotocal | Nautwanhila | Eosinophils | Pasanhila | Lymphogra | tes Monocytes | Platelets | Mean PlateletIf | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject No. | Actual Date<br>and Time | Phase | (10^9/L) | (10^9/L) | (10^9/L) | (10^9/L) | (10^9/L) | (10^9/L) | Volume<br>(fL) | Unscheduled,<br>Reason |
| <subject id=""></subject> | <ddmmmy<br>YYY hh:mm</ddmmmy<br> | | xx | XX | xx | XX | XX | XX | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

16.2.1.8.4. Biochemistry (I)

| Subject No. | Actual Date and Time | Protocol Phase | AST<br>(IU/L) | ALT<br>(IU/L) | GGT<br>(IU/L) | LDH<br>(IU/L) | ALP<br>(IU/L) | CK<br>(IU/L) | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy hh="" mm="" yy=""></ddmmmyy> | | XX | XXX | XX | xx | XX | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.8.5. Biochemistry (II)

| Subject No. | Actual Date and Time | Protocol Phase | Creatinine<br>(mg/dL) | eGFR | Urea<br>(mg/dL) | Sodium<br>(mmol/L) | Potassium<br>(mmol/L) | Calcium<br>(mg/dL) | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy hh="" mm="" yy=""></ddmmmyy> | <protocol<br>Phase&gt;</protocol<br> | XX | xxx | XX | xx | XX | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

16.2.1.8.6. Biochemistry (III)

| Subject No. | Actual Date and Time | Protocol Phase | Magnesium<br>(mg/dL) | Glucose<br>(mg/dL) | Total<br>Cholesterol<br>(mg/dL) | Triglycerides (mg/dL) | Albumin<br>(g/dL) | Total Protein<br>(g/dL) | If<br>Unscheduled<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy hh="" mm="" yy=""></ddmmmyy> | <protocol phase=""></protocol> | XX | XXX | XX | xx | XX | XX | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Version: <Version> Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.8.7. Biochemistry (IV)

| Subject No. | Actual Date<br>and Time | Protocol Phase | Uric Acid<br>(mg/dL) | Total Bilirubin<br>(mg/dL) | Direct<br>Bilirubin<br>(mg/dL) | Indirect<br>Bilirubin<br>(mg/dL) | TSH<br>(mIU/L) | Chloride<br>(mmol/L) | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy< td=""><td><protocol< td=""><td>XX</td><td>XXX</td><td>xx</td><td>XX</td><td>XX</td><td>XX</td><td><reason></reason></td></protocol<></td></ddmmmyy<> | <protocol< td=""><td>XX</td><td>XXX</td><td>xx</td><td>XX</td><td>XX</td><td>XX</td><td><reason></reason></td></protocol<> | XX | XXX | xx | XX | XX | XX | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Version: <Version> Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.8.8. Biochemistry (V)

| Subject No. | Actual Date and Time | Protocol Phase | Amylase<br>(g/dL) | LDL<br>Cholesterol<br>(mg/dL) | HDL<br>Cholesterol<br>(mg/dL) | FSH<br>(mg/dL) | C-Reactive<br>Protein | Cystain C | If<br>Unscheduled<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyy< td=""><td><protocol phase=""></protocol></td><td>XX</td><td>xxx</td><td>xx</td><td>XX</td><td>XX</td><td>xx</td><td><reason></reason></td></ddmmmyy<> | <protocol phase=""></protocol> | XX | xxx | xx | XX | XX | xx | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Version: <Version> Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

## 16.2.1.8.9. Coagulation

| Subject No. | Actual Date and<br>Time | Protocol Phase | Prothrombin Rate<br>(%) | Prothrombin<br>(sec) | Time INR | aPTT<br>(sec) | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <protocol phase=""></protocol> | XX | XX.X | x.xx | XX.X | <reason></reason> |

# <Insert as many rows as deemed necessary>

INR - International Normalized Ratio; aPTT - Activated Partial Thromboplastin Time

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

16.2.1.8.10. Urinalysis

| Subject<br>No. | Actual<br>Date and<br>Time | Protocol<br>Phase pH | Specific<br>Gravity | Protein | Hemoglobin | Glucose | Ketones | Bilirubin | Nitrites | | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <subject< td=""><td><ddmm<br>MYYYY<br/>hh:mm&gt;</ddmm<br></td><td><protoco<br>1 Phase&gt; xx x</protoco<br></td><td>x.xxx</td><td><qualitative<br>Value&gt;</qualitative<br></td><td><qualitative<br>Value&gt;</qualitative<br></td><td><qualitative<br>Value&gt;</qualitative<br></td><td><qualitative<br>Value&gt;</qualitative<br></td><td><qualitative<br>Value&gt;</qualitative<br></td><td><qualitative<br>Value&gt;</qualitative<br></td><td><qualitative<br>Value&gt;</qualitative<br></td><td><reason></reason></td></subject<> | <ddmm<br>MYYYY<br/>hh:mm&gt;</ddmm<br> | <protoco<br>1 Phase&gt; xx x</protoco<br> | x.xxx | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <qualitative<br>Value&gt;</qualitative<br> | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; NCR - Not Clinically Relevant; CR - Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.8.11. Urine Microscopy

| Subject No. | Actual Date and<br>Time | Protocol Phase | Squamous<br>Epithelial Cells<br>(/uL) | Erythrocytes<br>(/uL) | Leukocytes<br>(/uL) | Observations | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <protocol phase=""></protocol> | <qualitative<br>Value&gt;</qualitative<br> | xx | xx | <observations></observations> | <reason></reason> |

<Insert as many rows as deemed necessary>

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant; RU - Relevance Unknown

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.8.12. Pregnancy Test

| Subject No. | Actual Date and Time | Protocol Phase | Matrix | Result | If Unscheduled,<br>Reason |
|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy<br>hh:nm&gt;</ddmmmyyyy<br> | <protocol phase=""></protocol> | <serum or="" urine=""></serum> | <positive negative="" or=""></positive> | <reason></reason> |

<Insert as many rows as deemed necessary>

Program: SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.8.13. Additional (Not Planned) Laboratory Safety Tests

| Subject No. | Actual Date and<br>Time | Protocol Phase | Investigational<br>Product | Parameter | Results | Reason |
|---|---|---|---|---|---|---|
| <subject id=""></subject> | <ddmmmyyyy hh="" mm=""></ddmmmyyyy> | <protocol phase=""></protocol> | <investigational<br>Product&gt;</investigational<br> | <parameter></parameter> | <results></results> | <reason></reason> |

Program: <SAS Program>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

16.2.1.9. Vital Signs

| Subject No. | Scheduled<br>Time | Actual Date<br>and Time | Protocol<br>Phase | Investigation<br>Product | al SBP<br>(mmHg) | DBP<br>(mmHg) | Pulse Rate<br>(beats/min) | Body<br>Temperature<br>(°C) | Respiratory<br>Rate<br>(beats/min) | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | | YYY hh:mm> | | <investigation 1="" product=""></investigation> | na xx | XX | XX | XX | XX | <reason></reason> |

<Insert as many rows as deemed necessary>

SBP - Systolic Blood Pressure; DBP - Diastolic Blood Pressure

L - Low; H - High; CR - Clinically Relevant; NCR - Not Clinically Relevant

Program: <SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.10. 12-Lead ECG

| Subject No. | Scheduled<br>Time | Actual Date<br>and Time | Protocol Phase | Investigational<br>Product | QTcF<br>(msec) | Result | If Abnormal,<br>Reason | If Abnormal,<br>Clinically<br>Significant? | If<br>Unscheduled,<br>Reason |
|---|---|---|---|---|---|---|---|---|---|
| <subject id=""></subject> | <scheduled<br>Time or<br/>Unscheduled&gt;</scheduled<br> | <ddmmmyy<br>YY hh:mm&gt;</ddmmmyy<br> | <protocol<br>Phase&gt;</protocol<br> | <investigationa<br>Product&gt;</investigationa<br> | lxxx | <abnormal <br="">Normal&gt;</abnormal> | <reason for<br="">being<br/>considered<br/>abnormal&gt;</reason> | <yes no=""></yes> | <reason></reason> |

Insert as many rows as deemed necessary

Program: SAS Program>

Execution Date/Time: <ddMMMyyyy HH:MM>

Version: <Version> Date: <DDMMMYYYY>



Clinical Study Report ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# 16.2.1.11. Urine Sampling

| Subject No. | Day of Dose | Protocol Time | Col | lection Time | —Urine Volume |
|---|---|---|---|---|---|
| Subject No. | Day of Dose | Trotocor Time | Start | End | |
| <subject id=""></subject> | <day #=""></day> | <protocol time=""></protocol> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <ddmmmyyyy<br>hh:mm&gt;</ddmmmyyyy<br> | <abnormal normal=""></abnormal> |
| <insert as="" many="" row<="" td=""><td>vs as deemed necessary&gt;</td><td></td><td></td><td></td><td></td></insert> | vs as deemed necessary> | | | | |

Program: <SAS Program>
Execution Date/Time: <ddM/MMyyyy HH:MM>

# 14. ANNEXES

Annex 5: Data Blind Review Process Minute - Part 3

Annex 6: List of Subjects Dosed - Part 3

Statistical Analysis Plan ITF2357/Givinostat 10 mg/mL oral suspension EudraCT No: 2021-005756-11

# - Part 3: eight (8) subjects

Each subject will participate in one study part only.

### 5.3.1. Part 3

A sample size of 8 subjects will be enrolled. The sample size was determined by practical considerations and not based on statistical power calculations.

#### 5.4. Randomization

This is a fixed sequence study. Randomization is not applicable.

### 5.5. Blinding

The study will be conducted as open label. Blinding procedures are not applicable.

#### 6. STUDY ASSESSMENTS

For each study part, a summary of procedures for study assessments are presented in Section 2 of the CSP (Study Flow-Chart and Study Design Diagram) [1].

### 6.1. Safety Assessments

Subjects' safety will be monitored during the study.

Safety assessments will include pre-study medical history, physical examination, vital signs, 12-lead ECG, clinical laboratory tests and adverse event (AE) monitoring. Additional safety measurements may be performed at the discretion of the investigator for reasons related to subject safety.

Medications will be mentioned according to the World Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) classification system.

### 6.1.1. Medical History

Medical history will cover all relevant past or present information related to subject's health at the time of informed consent signature.

Medical history at screening will include past or present relevant cardiovascular, respiratory, renal, genitourinary, gastrointestinal, hepatic, hematological, immunological, endocrine, dermatological, musculoskeletal, neurological, psychiatric, drug and surgical history, or any other diseases or disorders.

Medical history will be referred in accordance with the Medical Dictionary for Regulatory Activities (MedDRA), version 24.1 or higher.

Adverse events related to medical history will be identified.

# 6.1.2. Physical Examination

Physical examination at screening and end-of-study will include: general appearance; skin; head and neck; thorax and abdomen; pulmonary auscultation; cardiac auscultation; abdomen palpation; limbs; brief neurological examination.

# 6.1.3. Weight, Height and Body Mass Index

The body height and weight values as well as the body mass index (BMI) will be recorded in the electronic case report form (eCRF) and will be determined at Screening. Only body weight will be determined also at admission and end-of-study.

The subjects' body weight will preferably be measured using the same weighing scale for all subjects and throughout the study. The weighing scale should have a precision of at least 0.5 kg.

# 6.1.4. Vital Signs

Vital signs will include:

- Systolic blood pressure (SBP).
- Diastolic blood pressure (DBP).
- Pulse rate (PR).
- Respiratory rate (RR).
- Body temperature.

# 6.1.5. 12 Lead Electrocardiogram

A 12-lead ECG will be performed preferably before the blood collection. The corrected QT interval by Fridericia (QTcF) will be analyzed.

# 6.1.6. Laboratory Safety Tests

The following laboratory parameters will be tested:

- Hematology:
  - Red blood cell (RBC) count.
  - White blood cell (WBC) count.
  - WBC differential count:
    - Neutrophils.
    - Eosinophils.
    - Basophils.
    - Lymphocytes.
    - Monocytes.
  - Hemoglobin.
  - Mean corpuscular volume (MCV).
  - Mean corpuscular hemoglobin (MCH).
  - Mean corpuscular hemoglobin concentration (MCHC).
  - Coefficient variation of the red cell distribution width (RDW-CV).
  - Hematocrit.
  - Platelet count.
  - Mean platelet volume.

- Specific gravity.
- Protein.
- Hemoglobin.
- Glucose.
- Ketones.
- Bilimbin
- Nitrites.
- Urobilinogen.
- Microscopy.
- Drugs-of-abuse urine test:
  - Cannabinoids.
  - Opiates.
  - Cocaine.
  - Amphetamines.
  - Benzodiazepines.
- Ethanol urine test.
- Cotinine urine test.
- Follicle-stimulating hormone (FSH) test.
- Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) diagnostic tests.

# 6.1.7. Adverse Events

The occurrence of clinical AEs will be monitored throughout the study.

Clinically significant abnormalities in laboratory safety tests, vital signs and physical examination will be reported as AEs.

Treatment-emergent AEs (TEAEs) are defined as AEs not present prior to first administration of investigational product, or AEs present before first administration of investigational product that worsen after the subject receives the first dose of investigational product. TEAEs that occur after administration of investigational product during the washout of a given period will be assigned to the treatment administered in that period.

The following information will be used for the description of the AEs:

- Reported Term.
- Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) coding.
- MedDRA Preferred Term (PT) coding.
- Start date and time.
- End date and time.
- Seriousness.
- Severity:
  - Mild.
  - Moderate.
  - Severe.
- Relationship (causality) for each treatment administrated, per part.
  - Reasonably Possible.
  - Not Reasonably Possible.
  - Unknown.

- Action taken:
  - Dose Increased.
  - Dose Not Changed.
  - Dose Rate Reduced.
  - Dose Reduced.
  - Drug Interrupted.
  - Drug Withdrawn.
  - Not Applicable.
  - Unknown.
- Concomitant medication.
- Outcome:
  - Fatal.
  - Not Recovered / Not Resolved.
  - Recovered / Resolved.
  - Recovered / Resolved with Sequelae.
  - Recovering / Resolving.
  - Unknown.
- Most recent study treatment taken.
- Last dosing date.

#### 6.1.8. Previous and Concomitant Medications

A previous medication is any medication for which the end date is prior to first dosing. A concomitant medication is any medication ongoing or initiated after first dosing.

For all study parts, the use of any medications including Over-the-Counter (OTC) products (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) is forbidden from 28 days or within 5 half-lives of the medicinal product, whichever is longer, prior to admission up to last sample for pharmacokinetics assessment, except for medications for the treatment of AEs.

Any medication (previous or concomitant) taken within the period of medication restriction must be recorded in the eCRF. If concomitant medication is ongoing at the follow-up visit, no end date will be provided in the eCRF.

For each study part, previous and concomitant medications used by study participants during the study and their judged impact on the pharmacokinetic assessment will be listed in the respective Data Blind Review Meeting/ Process Minute (Annex 5).

Concomitant medications will be coded according to the WHO ATC classification system.

#### 6.2. Pharmacokinetic Assessments

# 6.2.1. Blood Sampling for Pharmacokinetic Assessments

In each study part, while subject is confined at the clinical research unit, blood samples will be taken preferably via an indwelling cannula placed in a vein of an upper limb of the subject. During ambulatory visits, blood samples will be taken by direct venipuncture.

The actual time of all pharmacokinetic blood draws will be recorded and reported for all subjects. The pre-dose blood sample will be collected within 30 minutes before dosing. The post-dose blood samples will be collected within ±3 minutes from the scheduled sampling time. Greater deviations will be reported as a protocol deviation and its cause will be recorded.

In case blood sampling for pharmacokinetics and other procedures coincide in time, blood draws will have priority unless other procedures are necessary for assuring subject's safety.

will carry out the determination of plasma levels of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563), midazolam, 1-hydroxymidazolam and total and free dabigatran in accordance with the applicable principles of Good Laboratory Practices (GLP), using a previously validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) analytical method.

The planned lower limit of quantification (LLOQ) and upper limit of quantification (ULOQ) for:

- givinostat are 1 and 100 ng/mL.
- givinostat metabolite ITF2374 are 1 and 100 ng/mL.
- givinostat metabolite ITF2375 are 1 and 100 ng/mL.
- givinostat metabolite ITF2440 are 10 and 500 ng/mL.
- givinostat metabolite ITF2563 are 2 and 125 ng/mL.
- midazolam are 100 and 100000 pg/mL.
- 1-hydroxymidazolam are 100 and 50000 pg/mL.
- total dabigatran are 1 and 400 ng/mL.
- free dabigatran are 1 and 400 ng/mL.

LLOQ represents a value lower than or equal to 1/20 of estimated C<sub>max</sub> value. Any adjustment to this range will be documented in the study specific Bioanalytical Report, which will supersede the indicated range.

#### 6.2.1.1. Part 3

A total of forty-eight (48) blood samples will be collected as follows:

- Twenty-two (22) blood samples of 6 mL each will be collected in sodium heparin tubes at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60, 72, 84 and 96 hours after the administration of givinostat, on Days 1 and 13, for the determination of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) plasma concentrations.
- Four (4) blood samples of 6 mL each will be collected in sodium heparin tubes before the morning dose of givinostat on Days 9, 10, 11 and 12, for the determination of pre-dose (Ctrough) plasma concentration of givinostat and metabolites.

#### 6.2.2. Urine Sampling for Pharmacokinetic Assessments

#### 6.2.2.1. Part 3

Urine will be collected on Day -1 (baseline) and in the following intervals, on Days 1 and 13, for the determination of the amounts of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) excreted in urine: 0-12, 12-24, 24-36, 36-48, 48-72 and 72-96 post-dose.

The date and actual time of urine collection start and completion will be recorded and reported for all subjects.

will carry out the determination of urine levels of givinostat and its metabolites (ITF2374, ITF2375, ITF2440 and ITF2563) in accordance with the applicable principles of GLP using a previously validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) analytical method.

The planned lower limit of quantification (LLOQ) and upper limit of quantification (ULOQ) for:

- givinostat are 10 and 2500 ng/mL.
- givinostat metabolite ITF2374 are 5 and 2500 ng/mL.
- givinostat metabolite ITF2375 are 4 and 800 ng/mL.
- givinostat metabolite ITF2440 are 150 and 25000 ng/mL.
- givinostat metabolite ITF2563 are 10 and 5000 ng/mL.

# 6.2.3. Plasma Pharmacokinetic Parameters

The following pharmacokinetic parameters will be derived by standard non-compartmental analysis (NCA) methods from the single-dose plasma concentration versus time profiles, for:

- Part 3 (Day 1):
  - givinostat.
  - givinostat metabolites (ITF2374, ITF2375, ITF2440 and ITF2563).

| Parameter | Description |
|---|---|
| C <sub>max</sub> | Maximum observed concentration, directly obtained from the observed concentration versus time profile. |
| Tmax | Time of occurrence of maximum observed concentration. |
| AUC <sub>0-t</sub> <sup>1</sup> | Area under the concentration <i>versus</i> time curve (AUC) from time of dosing (t=0h) to the time of the last measurable concentration (t <sub>last</sub> ), calculated by the linear-up/log-down trapezoidal method. |
| $AUC_{0\text{-}\infty}$ | Total AUC extrapolated to infinity, calculated as $AUC_{0-t} + \frac{C_{last}}{\lambda_z}$ , where $C_{last}$ |
| | is the last measurable concentration and $\lambda_z$ is the apparent terminal elimination rate constant. |
| %AUC <sub>extrap</sub> | Percentage of AUC <sub>0-∞</sub> due to extrapolation from the time of the last measurable concentration ( $t_{last}$ ) to infinity, i.e., residual area, calculated as $100 \cdot \frac{AUC_{0-\infty} - AUC_{0-t}}{AUC_{0-\infty}}$ . |
| $\lambda_z$ | Apparent first order elimination rate constant associated with the terminal (log-linear) portion of the concentration <i>versus</i> time curve. The parameter is estimated by linear least square regression analysis using the last three (or more) non-zero concentrations. |
| t <sub>½</sub> | Apparent terminal elimination half-life, calculated as $\frac{ln(2)}{\lambda_2}$ . |

In Part 3, for givinostat and its metabolites the last sampling time corresponds to 96 hours.

In estimating the pharmacokinetic parameters, concentrations below the LLOQ before Tmax will be set to zero. After Tmax, concentrations below the LLOQ will be considered as missing. However, in case of two or more consecutive concentrations below the LLOQ, the first value will be replaced by 1/2 of the LLOQ value and the next values will be considered as missing.

Additional pharmacokinetic parameters may be calculated for the plasma concentration versus time profiles, if considered appropriate and justified at the time of the pharmacokinetic analysis.

#### 6.2.4. Urinary Pharmacokinetic Parameters

The following pharmacokinetic parameters will be derived by standard NCA methods from the urine excretion profiles, for the first dose (Day 1, single-dose) and the last dose (Day 13, multiple-dose):

- Part 3:
  - givinostat.
  - givinostat metabolites (ITF2374, ITF2375, ITF2440 and ITF2563).

| Parameter | Description |
|---|---|
| R <sub>max</sub> | Maximum observed urinary excretion rate. |
| tu <sub>max</sub> | Time of occurrence of maximum urinary excretion rate. |
| Amt <sub>CUM</sub> | Cumulative amount of drug excreted in urine, calculated as $\sum (Concentration \cdot Volume)$ |
| AURC <sub>0-t</sub> | Area under the urine excretion rate curve from time zero to last measurable observed excretion rate. |
| REC% | Percentage of drug recovered in urine, calculated for givinostat as 100 · Amt <sub>CUM</sub> , and for givinostat metabolites as 100 · AMT <sub>CUM,Metabolie</sub> /MW <sub>Metabolite</sub> , where MW represents the molecular weight of the analyte. |
| | Note: For givinostat, MW is 421.49 g/mol; for ITF2374, MW is 405.49 g/mol; for ITF2375, MW is 406.47 g/mol; for ITF2440, MW is 257.33 g/mol; and for ITF2563, MW is 178.19 g/mol. |
| CL <sub>R</sub> /F | Apparent renal clearance affected by F, calculated as $\frac{Dose}{AURC_{0-1}}$ . |

#### 7. STUDY ENDPOINTS

#### 7.1. Primary

 Givinostat and its metabolites plasma and urine concentrations and thereof derived pharmacokinetic parameters following single and multiple oral doses of givinostat (Part 3).

#### 7.2. Secondary

 Incidence and severity of AEs; changes in vital signs, physical examination, ECG and clinical laboratory tests following administration of single- and multiple-doses of givinostat (Part 3).

#### 8. ANALYSIS POPULATIONS

The analysis populations are defined in accordance with the CSP [1].

For each study part, the subjects to be included in each analysis population will be reported in the respective Data Blind Review Process Minute (Annex 5).

For each study part, explanation of the reasons for exclusion of subjects from any analysis population will be provided in the respective Data Blind Review Process Minute (Annex 5) and in the CSR.

The list of subjects who complete each study part will be presented in Annex 6.

#### 8.1. Part 3

# 8.1.1. Part 3 Safety Analysis Population

All subjects who receive at least one dose of the IMP in Part 3 of the study will constitute the Part 3 Safety Analysis Population.

Part 3 safety data analysis will be performed for all subjects in the Part 3 Safety Analysis Population.

### 8.1.2. Part 3 Pharmacokinetic Analysis Population

#### 8.1.2.1. Part 3 Single-Dose Pharmacokinetic Analysis Population

Part 3 Single-Dose Pharmacokinetic Analysis Population will include all subjects enrolled in Part 3 of the study, who are expected to provide evaluable pharmacokinetic data for the givinostat single-dose administration (Day 1), without deviations affecting pharmacokinetic interpretation.

The following reasons justify the exclusion of the pharmacokinetic data of a subject from the Part 3 single-dose pharmacokinetic analysis population:

 Protocol violation considered to have a potentially relevant effect on the pharmacokinetic results of the study.

NOTE: These protocol violations will be reported in the Data Blind Review Process Minute (Annex 5), and their impact will be assessed at the time of pharmacokinetic analysis.

Subject experienced vomiting or diarrhea.

NOTE: Subjects that experienced vomiting or diarrhoea during this study part will be reported in the Data Blind Review Process Minute (Annex 5), and their exclusion will be assessed at the time of pharmacokinetic analysis.

and/or SAS®.

In-text Tables and Figures will preferably be prepared in portrait format. Listings will preferably be prepared in landscape format.

The CSR will be written according to PPD SOPs and templates for reporting bioavailability/bioequivalence trials.

# 11.2. Planned Tables, Figures, and Subject Data Listings

The planned Tables, Figures, and Individual Data Listings for the CSR are listed below.

# 11.2.1. In-text Tables and Figures

For CSR Synopsis:

The following Tables will be produced for direct insertion in the Synopsis of the CSR:

| Title |
|---|
| PART 3 |
| Givinostat and Its Main Metabolites (ITF2374 and ITF2375,): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Plasma |
| Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| Givinostat and Its Main Metabolites (ITF2374 and ITF2375,): Summary Statistics of the Plasma Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Plasma |
| Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| Givinostat and Its Main Metabolites (ITF2374 and ITF2375): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Urinary |
| Pharmacokinetic Parameters Following Single-Dose Administration of Givinostat (Day 1) |
| Givinostat and Its Main Metabolites (ITF2374 and ITF2375): Summary Statistics of the Urinary Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |
| Givinostat Metabolites (ITF2440 and ITF2563): Summary Statistics of the Urinary |
| Pharmacokinetic Parameters Following Multiple-Dose Administration of Givinostat (Day 13) |

The following Figures will be produced for direct insertion in the Synopsis of the CSR:

| Lege | nd |
|---|---|
| PAR | T 3 |
| Givi | nostat: Geometric Mean (95% CI) Plasma Concentration Versus Time Profile Following<br>le-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat. A – Linear |

| In-text Figures | Legend |
|---|---|
| | Amount Urinary Excretion <i>Versus</i> Time Profile Following Single-Dose (Day 1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.J.1. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) of Urinary<br>Excretion <i>Versus</i> Time Profile Following Single-Dose (Day 1) and Multiple-<br>Dose (Day 13) Administration of Givinostat – Linear Scale |
| Figure 3.J.2. | Givinostat Metabolite (ITF2563): Geometric Mean (95% CI) of Cumulative<br>Amount Urinary Excretion <i>Versus</i> Time Profile Following Single-Dose (Day<br>1) and Multiple-Dose (Day 13) Administration of Givinostat – Linear Scale |

# 11.2.2. Tables, Figures and Graphs Referred to But Not Included in the Text (Section 14 of CSR)

At least the following Tables and Figures should be produced for Section 14 of the CSR. If necessary, additional Tables and Figures should be prepared.

The following Tables and Figures will be compiled in a document, to be considered as Section 14 (Tables, Figures and Graph Referred To But Not Included in the Text) of the CSR.

| End-of-Text<br>Tables | Title |
|---|---|
| 14.3. PART 3 | Transfer and the second of the |
| 14.3.1. DEMOC | GRAPHIC DATA – PART 3 |
| 14.3.1.1. | Demographic Data – Part 3 Safety Analysis Population |
| 14.3.1.2. | Demographic Data – Part 3 Single-Dose Pharmacokinetic Analysis<br>Population |
| 14.3.1.3. | Demographic Data – Part 3 Multiple-Dose Pharmacokinetic Analysis<br>Population |
| 14.3.1.4. | Subjects Prematurely Discontinued After First Dosing |
| 14.3.2. PHARM | IACOKINETIC DATA – PART 3 |
| 14.3.2.1. | Plasma Pharmacokinetic Data |
| 14.3.2.1.1. | Deviations from Blood Sampling Schedule |
| 14.3.2.1.1.1. | Deviations from Blood Sampling Schedule |
| 14.3.2.1.1.2. | Missing Blood Samples |
| 14.3.2.1.1.3. | Other Important Protocol Deviations |
| 14.3.2.1.2. | Plasma Concentrations |
| 14.3.2.1.2.1. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Concentrations Following Single-Dose Administration of Givinostat (Day 1) |
| 14.3.2.1.2.2. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Concentrations Following Single-Dose Administration of Givinostat (Day 1)<br>– Male Subjects |
| 14.3.2.1.2.3. | Givinostat: Individual Data and Descriptive Statistics of Plasma<br>Concentrations Following Single-Dose Administration of Givinostat (Day 1)<br>- Female Subjects |
| 14.3.2.1.2.4. | Givinostat Metabolite (ITF2374): Individual Data and Descriptive Statistics of Plasma Concentrations Following Single-Dose Administration of Givinostat (Day 1) |



# 11.2.3. List of Subject Data Listings (Section 16.2 of CSR)

The following Data Listings will be produced for Section 16.2. Subject Data Listings of the CSR.

If necessary, additional Data Listings should be prepared.

| Listing No. | Title |
|---|---|
| 16.2. SUBJECT | TS DATA LISTING |
| 16.2.3. Part 3 | |
| 16.2.3.1. | Subject Disposition |
| 16.2.3.1.1. | Subject Disposition |
| 16.2.3.2. | Protocol Deviations |
| 16.2.3.2.1. | Blood Sampling Times Deviations |
| 16.2.3.2.2. | Other Protocol Deviations |
| 16.2.3.3. | Excluded Data from the Pharmacokinetic Analysis |
| 16.2.3.3.1. | Plasma Concentrations |
| 16.2.3.3.1.1. | Individual Data of Plasma Concentrations |
| 16.2.3.3.2. | Plasma Concentration Versus Time Profiles |
| 16.2.3.3.2.1. | Individual Plasma Concentration Versus Time Profiles - Linear Scale |
| 16.2.3.3.2.2. | Individual Plasma Concentration Versus Time Profiles - Semi-Logarithmic |
| | Scale |
| 16.2.3.3.3. | Urine Excretion |
| 16.2.3.3.3.1. | Individual Data of Plasma Concentrations |
| 16.2.3.3.4. | Urine Excretion Versus Time Profiles |
| 16.2.3.3.4.1. | Urine Excretion Versus Time Profiles – Linear Scale |
| 16.2.3.4. | Demographic and Other Baseline Data |
| 16.2.3.4.1. | Demographic Data |
| 16.2.3.4.2. | Fertility/Contraception |
| 16.2.3.4.2.1. | Female Fertility/Contraception |
| 16.2.3.4.2.2. | Male Fertility/Contraception |
| 16.2.3.4.3. | Drugs of Abuse, Ethanol and Cotinine |
| 16.2.3.4.4. | Viral Serology at Screening |
| 16.2.3.4.5. | Previous and Concomitant Medication |
| 16.2.3.4.6. | SARS-COV-2 Test |
| 16.2.3.5. | Compliance |
| 16.2.3.5.1. | Investigational Product Administration |
| 16.2.3.6. | Individual Pharmacokinetic Data |
| 16.2.3.6.1. | Givinostat: Individual Pharmacokinetic Data |
| 16.2.3.6.1.1. | Givinostat: Individual Drug Plasma Concentration Data |
| 16.2.3.6.1.2. | Givinostat: Individual Plasma Pharmacokinetic Parameters |
| 16.2.3.6.1.3. | Givinostat: Individual Plasma Pharmacokinetic Profiles |
| 16.2.3.6.1.4. | Givinostat: Individual Urine Excretion Data |
| 16.2.3.6.1.5. | Givinostat: Individual Urine Pharmacokinetic Parameters |
| 16.2.3.6.1.6. | Givinostat: Individual Urine Pharmacokinetic Profiles |
| 16.2.3.6.1.7. | Givinostat: Documentation of Statistical Analysis |
| 16.2.3.6.1.7.1. | Givinostat: Plasma Non-Compartmental Analysis Output |
| 16.2.3.6.1.7.2. | Givinostat: Plasma Non-Compartmental Analysis Plots |
| 16.2.3.6.1.7.3. | Givinostat: Urine Non-Compartmental Analysis Output |